



# CAR-T IMMUNOMONITORING DANS LE MYELOME MULTIPLE

# CART-I5M

# PROTOCOLE DE RECHERCHE INTERVENTIONNELLE IMPLIQUANT LA PERSONNE HUMAINE DE CATEGORIE 2 CONTRAINTES ET RISQUES MINIMES

Version n°2 du 08/10/2025 Numéro ID-RCB: 2025-A01924-45

Cette étude clinique a obtenu le financement de Intergroupe France Myélome et Sport et Collection

# **Promoteur:**

Centre Hospitalier Universitaire de Poitiers 2 rue de la Milétrie CS 90577 86021 POITIERS cedex Tél: 05 49 44 33 89

# **Investigateur coordonnateur:**

Dr BOBIN Arthur

Service d'Oncologie Hématologique et de Thérapie cellulaire Centre Hospitalier Universitaire de Poitiers 2 rue de la Milétrie – CS 90577 86021 Poitiers cedex Tél: 05 49 44 42 01

E-mail: arthur.bobin@chu-poitiers.fr

 $Ce\ protocole\ a\ \acute{e}t\acute{e}\ conçu\ et\ r\acute{e}dig\acute{e}\ \grave{a}\ partir\ de\ la\ version\ 4.0\ du\ 18/01/2022\ du\ protocole-type\ du\ GIRCI\ SOHO$ 

CE DOCUMENT CONFIDENTIEL EST LA PROPRIETE DU CHU DE POITIERS.

AUCUNE INFORMATION NON PUBLIEE FIGURANT DANS CE DOCUMENT NE PEUT ETRE DIVULGUEE SANS

AUTORISATION ECRITE PREALABLE DU CHU DE POITIERS

Version n°2 du 08.10.2025 CONFIDENTIEL Page 1 sur 54





# HISTORIQUE DES MISES A JOUR DU PROTOCOLE

| VERSION | DATE | RAISON DE LA MISE A JOUR |
|---------|------------|--------------------------|
| 1 | 25/08/2025 | Version initiale |
| 2 | 08/10/2025 | Commentaires CPP IDF IV |





# PAGE DE SIGNATURE DU PROTOCOLE

### SIGNATURE DU PROTOCOLE

# Signature de l'Investigateur Coordonnateur

Dr BOBIN Arthur

Date: 08.10.2025

Signature:

# Signature du Promoteur

Pour la Directrice Générale et par délégation La Directrice de la Recherche Emmanuelle DE LAVALETTE-FERGUSON

Date: 08.10.2025

Signature:







# PRINCIPAUX CORRESPONDANTS

**Investigateur coordonnateur/principal:** 

Dr BOBIN Arthur

Service d'Oncologie Hématologique et de Thérapie

cellulaire

Centre Hospitalier Universitaire de Poitiers

2 rue de la Milétrie CS 90577

86021 Poitiers cedex

Tél: 05 49 44 42 01

E-mail: arthur.bobin@chu-poitiers.fr

Promoteur:

Centre Hospitalier Universitaire de Poitiers

Direction de la Recherche

2 Rue de la Milétrie - CS 90577

86021 POITIERS Cedex Tél: 05 49 44 33 89

Email: drc.promointerne@chu-poitiers.fr

**Services Participants:** 

Service d'Oncologie Hématologique et de Thérapie Email : data-management@chu-poitiers.fr

cellulaire **CIC P1042**  **Data-Management:** 

<u>Autres spécialités :</u>

Groupe IRATI "ImmunoRégulation, Alarmines et

cellules T Innées"

**INSERM U1313-IRMETIST** 

Pôle Biologie Santé -Bâtiment B36

Aile A. 3ème étage. Secteur beta

1, rue Georges Bonnet BP 633

86022 Poitiers

Tél: 05 49 45 43 41

**Centre de Ressources Biologiques UF 9008 :** 

Centre Hospitalier Universitaire de Poitiers 5 cour Est -2 rue de la Milétrie -CS 90577

86021 Poitiers

Michèle GROSDENIER

Email: michele.grosdenier.bruneau@chu-poitiers.fr

Tél: 05 49 44 31 74

Responsables scientifiques:

Dr André HERBELIN

Pr Jean-Marc GOMBERT

Dr. Alice BARBARIN





# **SOMMAIRE**

| 1 | RESUM | E | 8 |
|---|---|---|---|
| 2 | JUSTIFI | CATION SCIENTIFIQUE ET DESCRIPTION GENERALE | 12 |
| | 2.1 | Etat actuel des connaissances | 12 |
| | 2.2 | Hypothèse de l'étude clinique et résultats attendus | 17 |
| | 2.3 | Bénéfices / risque | 18 |
| | 2.4 | Retombées attendues | 19 |
| | 2.5 | Justification recherche dénuée de risques | 19 |
| 3 | | TIFS ET CRITERE DE JUGEMENT PRINCIPAL | 21 |
| | 3.1 | Objectif principal : | 21 |
| | 3.2 | Critère de jugement principal : | 21 |
| 4 | | FIFS ET CRITERES DE JUGEMENT SECONDAIRES | 22 |
| • | 4.1 | Objectifs secondaires | 22 |
| | 4.2 | Critères de jugement secondaires | 22 |
| 5 | | LES D'ÉLIGIBILITE | 23 |
| J | 5.1 | Critères d'inclusion | 23 |
| | 5.2 | Critères de non-inclusion | 23 |
| | 5.3 | Faisabilités et modalités de recrutement | 23 |
| 6 | | PTION DE L'ETUDE CLINIQUE | 25 |
| U | 6.1 | Justification des choix méthodologiques | 25<br>25 |
| | 6.2 | • | 2 <i>5</i> |
| 7 | | Schéma de l'étude clinique | 26 |
| 7 | | LEMENT DE L'ETUDE | |
| | 7.1 | Calendrier Table on the spirit lastif to a printing and the spirit | 26<br>27 |
| | 7.2 | Tableau récapitulatif du suivi participant | 27 |
| | 7.3 | Visite de pré-inclusion/inclusion | 28 |
| | 7.4 | Visites de suivi | 29 |
| | 7.5 | Visite de fin | 30 |
| | 7.6 | Règles d'arrêt | 30 |
| | 7.7 | Contraintes liées à l'étude clinique et indemnisation éventuelle des participants | 31 |
| | 7.8 | Inscription du participant de l'étude clinique dans le fichier national des personnes qui se pr | |
| | | des recherches | 31 |
| 8 | | DURE ET STRATEGIES | 32 |
| | 8.1 | Analyse cellulaire des prélèvements de sang total et de moelle osseuse : | 32 |
| | 8.2 | Analyses supervisées : | 32 |
| | 8.3 | Analyses non supervisées : | 33 |
| | 8.4 | Dosages cytokiniques des sérums : | 33 |
| 9 | Colle | CTION D'ECHANTILLONS BIOLOGIQUES | 34 |
| | 9.1 | Description des collections | 34 |
| | 9.2 | Transports | 35 |
| | 9.3 | Conservation | 35 |
| | 9.4 | Devenir de la collection | 35 |
| 1( | O GESTIC | N DES EVENEMENTS INDESIRABLES / EFFETS INDESIRABLES / INCIDENTS | 37 |
| 11 | 1 ASPECT | TS STATISTIQUES | 38 |
| | 11.1 | Calcul de la taille d'étude | 38 |
| | 11.2 | Méthodes statistiques employées | 38 |
| 12 | 2 GESTIC | N ET TRAITEMENT DES DONNEES ET DOCUMENTS SOURCE | 39 |
| | 12.1 | Données et documents source | 39 |
| | 12.2 | Consignes pour le recueil des données | 39 |
| | 12.3 | Gestion et circuit des données | 40 |
| | 12.4 | Confidentialité des données | 40 |
| | 12.5 | Conservation des documents et des données relatifs à l'étude | 41 |
| | 12.6 | Cession des données | 41 |
| 13 | | OLE ET ASSURANCE QUALITE | 42 |
| | | | - |



# CART-I5M

| 13.1 | Accès aux données | 42 |
|---------|----------------------------------------------|----|
| 13.2 | Contrôle Qualité | 42 |
| 13.3 | Audit et inspections | 42 |
| 14 Cons | SIDERATIONS ETHIQUES ET REGLEMENTAIRES | 43 |
| 15 REGI | LES RELATIVES A LA PUBLICATION | 45 |
| 15.1 | Communications scientifiques | 45 |
| 15.2 | Communication des résultats aux participants | 45 |
| 16 Réfé | ÉRENCES BIBLIOGRAPHIQUES | 46 |
| ANNEXE | ES | 48 |

Version n°2 du 08.10.2025 CONFIDENTIEL Page **6** sur **54** 





# Liste des abréviations

Ac Anticorps

ANSM Agence Nationale de Sécurité du Médicament et des produits de santé

ARC Attaché de Recherche Clinique BCMA B-cell maturation antigen BiTEs bispecific - cell engagers

CAR-T chimeric antigen receptor T cell CPP Comité de Protection des Personnes

CRAB Calcium, renal failure, anemia, bone lesion

CRB Centre de Ressources Biologiques

CRF/e-CRF Case Report Form / Electronic Case Report Form

DMSO Diméthylsulfoxyde

EMRA Effector memory re-expressing CD45RA

Eomes Eomesodermin

ICH International Council for Harmonisation

IFN Interféron

Ig Immunoglobuline
IL Interleukine
iNKT Invariant NKT

KIR Killer inhibitor receptor

LT Lymphocyte T

LT- $\gamma\delta$  Lymphocytes T gamma delta

LTI Lymphocytes T innés

MAIT Mucosal-Associated Invariant T

MDSC Myeloid-derived suppressive cells; cellules myéloïdes suppressives

MEM Microenvironnement médullaire MFI Mean fluorescence intensity

MGUS Monoclonal gammapathy of undetermined/unknown significance; gammapathie de signification

indéterminée

MM Myélome multiple MO Moelle osseuse

MR Méthodologie de référence

MESR Ministère de l'Enseignement Supérieur et de la Recherche

NDMM Newly diagnosed multiple myeloma; myélome multiple nouvellement diagnostiqué

PBMC Peripheral blood mononuclear cell PLZF Promyelocytic Leukemia Zinc Finger

RGPD Règlement Général sur la Protection des Données

RRMM Relapsed/refractory multiple myeloma; myélome multiple en rechute/réfractaire

sMM smoldering multiple myeloma; myélome indolent/asymptomatique

T-Bet T-box expressed in T cells

TCR T Cell Receptor

TGF Transforming Growth Factor

TIGIT T cell immunoreceptor with Ig and ITIM domains
TIM-3 T cell immunoglobulin and mucin containing protein-3
TRM T resident memory; Lymphocytes T résidents mémoires





# 1 Résumé

Version n°2 du 08.10.2025 2025-A01924-45

| TITRE | CAR-T IMMunoMonitoring dans le Myelome Multiple –<br>CART-I5M |
|---|---|
| PROMOTEUR | Centre Hospitalier Universitaire de Poitiers<br>2 rue de la Milétrie – CS 90577<br>86021 Poitiers cedex<br>Tél: 05 49 44 33 89 |
| INVESTIGATEUR COORDONNATEUR/PRINCIPAL | Dr BOBIN Arthur Centre Hospitalier Universitaire de Poitiers Service d'Oncologie Hématologique et de Thérapie cellulaire 2 rue de la Milétrie – CS 90577 – 86021 Poitiers cedex Tél: 05 49 44 42 01 E-mail: arthur.bobin@chu-poitiers.fr |
| JUSTIFICATION / CONTEXTE | Le myélome multiple (MM) est une maladie incurable malgré les progrès thérapeutiques récents. Une des nouvelles thérapies consiste à utiliser des cellules CAR-T (chimeric antigen receptor T-cell), des lymphocytes T du patient modifiés pour exprimer un TCR transgénique ciblant la protéine BCMA présente à la surface des plasmocytes tumoraux. Cette stratégie, bien que coûteuse est efficace. Cependant, de nombreuses questions restent sans réponses, comme pouvoir prédire la persistance des CAR-T après réinjection chez le patient, leur effet bystander sur le système immunitaire du patient en reconstitution et en particulier la prise en compte de certains sous-types immunitaires comme les lymphocytes T innés (LTI), tels que les LT-γδ, MAIT, iNKT et LTI CD8. Nous émettons ici l'hypothèse que le caractère souche (ou <i>stemness</i> ) des LT avant l'aphérèse et son maintien après activation/stimulation peut prédire la persistance des LT CAR-BCMA chez le patient, un critère reconnu de la bonne réponse au traitement par cette thérapie. |
| OBJECTIF PRINCIPAL | Corrélation du caractère souche ou <i>stemness</i> , reflétée par l'expression du facteur de transcription TCF1, des lymphocytes T (CD3+) avant l'aphérèse destinée à la production du CAR-BCMA, avec : 1) la persistance des lymphocytes CAR-BCMA chez le patient, dans le sang périphérique aux différents temps du suivi longitudinal sur 1 an ; 2) la réponse à la thérapie CAR-T anti-BCMA. |
| CRITERES DE JUGEMENT<br>PRINCIPAL | 1) Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation avec le pourcentage de LT CAR-BCMA(+) aux différents temps de suivi sur un an. 2) Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation avec la profondeur de la réponse du patient telle que définie par les recommandations internationales (IMS/IMWG). |



CART-I5M

| | 1. Déterminer si le caractère souche ou stemness, reflété par |
|---|---|
| | l'expression du facteur de transcription TCF1, des lymphocytes T |
| | (CD3+) avant l'aphérèse et/ou la lymphodéplétion, est corrélé |
| | avec la persistance des lymphocytes CAR-BCMA chez le patient, |
| | dans la moelle osseuse à M3 et à M12. |
| | 2. Identifier les mécanismes d'homéostasie de la réponse immunitaire, |
| | reflétés par l'expression de CD95L membranaire et la |
| OBJECTIF SECONDAIRES | différenciation précoce (precocius differenciation), interférent avec |
| | la persistance des LT CAR-BCMA(+) dans le sang périphérique aux |
| | différents temps du suivi longitudinal sur 1 an. |
| | 3. Déterminer si le profil inflammatoire des patients, déterminé par |
| | dosages cytokiniques (sCD95L, IL-1β, IFN-γ, IL-6, IL-10, IL-15 |
| | TNF-α) à chaque temps est inversement corrélé avec la persistance |
| | des LT CAR-BCMA(+) en périphérie et/ou dans la moelle osseuse. |
| | Analyse longitudinale des pourcentages des LT conventionnels |
| | (CD4, Treg, CD8 et leurs différentes sous-populations) et non |
| | conventionnels (iNKT, LT-γδ, MAIT et LTI CD8) en périphérie et |
| | dans la moelle osseuse, dans les fractions CART-BCMA(+) et |
| | CART-BCMA(-) et analyse des critères suivants : |
| | - Expression de CD95 et CD95L membranaire, |
| | - État d'exhaustion : expression des marqueurs PD-1, TIM-3, |
| | TIGIT, LAG-3, |
| | - Arsenal cytotoxique : expression de perforine et de |
| | granzymes, |
| CRITERES DE JUGEMENT | - Signatures transcriptionnelles : facteurs de transcription |
| SECONDAIRES | Homes I-bet Helios PL/H |
| SECONDAIRES | Eomes, T-bet, Helios, PLZF. Niveau d'expression du facteur de transcription TCF-1 (MFI) dans |
| SECONDAIRES | 2. Niveau d'expression du facteur de transcription TCF-1 (MFI) dans |
| SECONDAIRES | 2. Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation |
| SECONDAIRES | 2. Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation avec la persistance des LT CART-BCMA (mesurée par le |
| SECONDAIRES | 2. Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation avec la persistance des LT CART-BCMA (mesurée par le pourcentage de LT CAR-BCMA(+)) dans la moelle osseuse à M3 et |
| SECONDAIRES | 2. Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation avec la persistance des LT CART-BCMA (mesurée par le pourcentage de LT CAR-BCMA(+)) dans la moelle osseuse à M3 et à M12. |
| SECONDAIRES | <ol> <li>Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation avec la persistance des LT CART-BCMA (mesurée par le pourcentage de LT CAR-BCMA(+)) dans la moelle osseuse à M3 et à M12.</li> <li>Mesure des concentrations de cytokines (sCD95L, IL-1β, IFN-γ, IL-</li> </ol> |
| SECONDAIRES | <ol> <li>Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation avec la persistance des LT CART-BCMA (mesurée par le pourcentage de LT CAR-BCMA(+)) dans la moelle osseuse à M3 et à M12.</li> <li>Mesure des concentrations de cytokines (sCD95L, IL-1β, IFN-γ, IL-6, IL-10, IL-15 et TNF-α) dans le sérum des patients avant aphérèse</li> </ol> |
| SECONDAIRES | <ol> <li>Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation avec la persistance des LT CART-BCMA (mesurée par le pourcentage de LT CAR-BCMA(+)) dans la moelle osseuse à M3 et à M12.</li> <li>Mesure des concentrations de cytokines (sCD95L, IL-1β, IFN-γ, IL-6, IL-10, IL-15 et TNF-α) dans le sérum des patients avant aphérèse et à chaque temps après injection du produit CART-BCMA et</li> </ol> |
| SECONDAIRES | <ol> <li>Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation avec la persistance des LT CART-BCMA (mesurée par le pourcentage de LT CAR-BCMA(+)) dans la moelle osseuse à M3 et à M12.</li> <li>Mesure des concentrations de cytokines (sCD95L, IL-1β, IFN-γ, IL-6, IL-10, IL-15 et TNF-α) dans le sérum des patients avant aphérèse et à chaque temps après injection du produit CART-BCMA et corrélation avec le pourcentage de LT CAR-BCMA(+) des LT</li> </ol> |
| SECONDAIRES | <ol> <li>Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation avec la persistance des LT CART-BCMA (mesurée par le pourcentage de LT CAR-BCMA(+)) dans la moelle osseuse à M3 et à M12.</li> <li>Mesure des concentrations de cytokines (sCD95L, IL-1β, IFN-γ, IL-6, IL-10, IL-15 et TNF-α) dans le sérum des patients avant aphérèse et à chaque temps après injection du produit CART-BCMA et corrélation avec le pourcentage de LT CAR-BCMA(+) des LT CAR-BCMA(+) en périphérie et/ou dans la moelle osseuse.</li> </ol> |
| SECONDAIRES | <ol> <li>Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation avec la persistance des LT CART-BCMA (mesurée par le pourcentage de LT CAR-BCMA(+)) dans la moelle osseuse à M3 et à M12.</li> <li>Mesure des concentrations de cytokines (sCD95L, IL-1β, IFN-γ, IL-6, IL-10, IL-15 et TNF-α) dans le sérum des patients avant aphérèse et à chaque temps après injection du produit CART-BCMA et corrélation avec le pourcentage de LT CAR-BCMA(+) des LT CAR-BCMA(+) en périphérie et/ou dans la moelle osseuse.</li> <li>Il s'agit d'une étude prospective interventionnelle avec risques et</li> </ol> |
| SECONDAIRES | <ol> <li>Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation avec la persistance des LT CART-BCMA (mesurée par le pourcentage de LT CAR-BCMA(+)) dans la moelle osseuse à M3 et à M12.</li> <li>Mesure des concentrations de cytokines (sCD95L, IL-1β, IFN-γ, IL-6, IL-10, IL-15 et TNF-α) dans le sérum des patients avant aphérèse et à chaque temps après injection du produit CART-BCMA et corrélation avec le pourcentage de LT CAR-BCMA(+) des LT CAR-BCMA(+) en périphérie et/ou dans la moelle osseuse.</li> <li>Il s'agit d'une étude prospective interventionnelle avec risques et contraintes minimes de catégorie 2, descriptive Exploratoire,</li> </ol> |
| SCHEMA DE L'ETUDE CLINIQUE | <ol> <li>Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation avec la persistance des LT CART-BCMA (mesurée par le pourcentage de LT CAR-BCMA(+)) dans la moelle osseuse à M3 et à M12.</li> <li>Mesure des concentrations de cytokines (sCD95L, IL-1β, IFN-γ, IL-6, IL-10, IL-15 et TNF-α) dans le sérum des patients avant aphérèse et à chaque temps après injection du produit CART-BCMA et corrélation avec le pourcentage de LT CAR-BCMA(+) des LT CAR-BCMA(+) en périphérie et/ou dans la moelle osseuse.</li> <li>Il s'agit d'une étude prospective interventionnelle avec risques et contraintes minimes de catégorie 2, descriptive Exploratoire,</li> <li>Non randomisée,</li> </ol> |
| | <ol> <li>Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation avec la persistance des LT CART-BCMA (mesurée par le pourcentage de LT CAR-BCMA(+)) dans la moelle osseuse à M3 et à M12.</li> <li>Mesure des concentrations de cytokines (sCD95L, IL-1β, IFN-γ, IL-6, IL-10, IL-15 et TNF-α) dans le sérum des patients avant aphérèse et à chaque temps après injection du produit CART-BCMA et corrélation avec le pourcentage de LT CAR-BCMA(+) des LT CAR-BCMA(+) en périphérie et/ou dans la moelle osseuse.</li> <li>Il s'agit d'une étude prospective interventionnelle avec risques et contraintes minimes de catégorie 2, descriptive Exploratoire, <ul> <li>Non randomisée,</li> <li>Longitudinale,</li> </ul> </li> </ol> |
| | <ol> <li>Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation avec la persistance des LT CART-BCMA (mesurée par le pourcentage de LT CAR-BCMA(+)) dans la moelle osseuse à M3 et à M12.</li> <li>Mesure des concentrations de cytokines (sCD95L, IL-1β, IFN-γ, IL-6, IL-10, IL-15 et TNF-α) dans le sérum des patients avant aphérèse et à chaque temps après injection du produit CART-BCMA et corrélation avec le pourcentage de LT CAR-BCMA(+) des LT CAR-BCMA(+) en périphérie et/ou dans la moelle osseuse.</li> <li>Il s'agit d'une étude prospective interventionnelle avec risques et contraintes minimes de catégorie 2, descriptive Exploratoire, <ul> <li>Non randomisée,</li> <li>Longitudinale,</li> <li>Monocentrique,</li> </ul> </li> </ol> |
| | <ol> <li>Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation avec la persistance des LT CART-BCMA (mesurée par le pourcentage de LT CAR-BCMA(+)) dans la moelle osseuse à M3 et à M12.</li> <li>Mesure des concentrations de cytokines (sCD95L, IL-1β, IFN-γ, IL-6, IL-10, IL-15 et TNF-α) dans le sérum des patients avant aphérèse et à chaque temps après injection du produit CART-BCMA et corrélation avec le pourcentage de LT CAR-BCMA(+) des LT CAR-BCMA(+) en périphérie et/ou dans la moelle osseuse.</li> <li>Il s'agit d'une étude prospective interventionnelle avec risques et contraintes minimes de catégorie 2, descriptive Exploratoire, <ul> <li>Non randomisée,</li> <li>Longitudinale,</li> <li>Monocentrique,</li> <li>A visée fondamentale.</li> </ul> </li> </ol> |
| | <ol> <li>Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation avec la persistance des LT CART-BCMA (mesurée par le pourcentage de LT CAR-BCMA(+)) dans la moelle osseuse à M3 et à M12.</li> <li>Mesure des concentrations de cytokines (sCD95L, IL-1β, IFN-γ, IL-6, IL-10, IL-15 et TNF-α) dans le sérum des patients avant aphérèse et à chaque temps après injection du produit CART-BCMA et corrélation avec le pourcentage de LT CAR-BCMA(+) des LT CAR-BCMA(+) en périphérie et/ou dans la moelle osseuse.</li> <li>Il s'agit d'une étude prospective interventionnelle avec risques et contraintes minimes de catégorie 2, descriptive Exploratoire, <ul> <li>Non randomisée,</li> <li>Longitudinale,</li> <li>Monocentrique,</li> <li>A visée fondamentale.</li> </ul> </li> <li>Tous les patients inclus dans cette recherche devront vérifier tous les</li> </ol> |
| | <ol> <li>Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation avec la persistance des LT CART-BCMA (mesurée par le pourcentage de LT CAR-BCMA(+)) dans la moelle osseuse à M3 et à M12.</li> <li>Mesure des concentrations de cytokines (sCD95L, IL-1β, IFN-γ, IL-6, IL-10, IL-15 et TNF-α) dans le sérum des patients avant aphérèse et à chaque temps après injection du produit CART-BCMA et corrélation avec le pourcentage de LT CAR-BCMA(+) des LT CAR-BCMA(+) en périphérie et/ou dans la moelle osseuse.</li> <li>Il s'agit d'une étude prospective interventionnelle avec risques et contraintes minimes de catégorie 2, descriptive Exploratoire, <ul> <li>Non randomisée,</li> <li>Longitudinale,</li> <li>Monocentrique,</li> <li>A visée fondamentale.</li> </ul> </li> <li>Tous les patients inclus dans cette recherche devront vérifier tous les critères d'inclusion listés ci-dessous :</li> </ol> |
| | <ol> <li>Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation avec la persistance des LT CART-BCMA (mesurée par le pourcentage de LT CAR-BCMA(+)) dans la moelle osseuse à M3 et à M12.</li> <li>Mesure des concentrations de cytokines (sCD95L, IL-1β, IFN-γ, IL-6, IL-10, IL-15 et TNF-α) dans le sérum des patients avant aphérèse et à chaque temps après injection du produit CART-BCMA et corrélation avec le pourcentage de LT CAR-BCMA(+) des LT CAR-BCMA(+) en périphérie et/ou dans la moelle osseuse.</li> <li>Il s'agit d'une étude prospective interventionnelle avec risques et contraintes minimes de catégorie 2, descriptive Exploratoire, <ul> <li>Non randomisée,</li> <li>Longitudinale,</li> <li>Monocentrique,</li> <li>A visée fondamentale.</li> </ul> </li> <li>Tous les patients inclus dans cette recherche devront vérifier tous les critères d'inclusion listés ci-dessous : <ul> <li>Consentement écrit donné par le participant,</li> </ul> </li> </ol> |
| SCHEMA DE L'ETUDE CLINIQUE | <ol> <li>Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation avec la persistance des LT CART-BCMA (mesurée par le pourcentage de LT CAR-BCMA(+)) dans la moelle osseuse à M3 et à M12.</li> <li>Mesure des concentrations de cytokines (sCD95L, IL-1β, IFN-γ, IL-6, IL-10, IL-15 et TNF-α) dans le sérum des patients avant aphérèse et à chaque temps après injection du produit CART-BCMA et corrélation avec le pourcentage de LT CAR-BCMA(+) des LT CAR-BCMA(+) en périphérie et/ou dans la moelle osseuse.</li> <li>Il s'agit d'une étude prospective interventionnelle avec risques et contraintes minimes de catégorie 2, descriptive Exploratoire, <ul> <li>Non randomisée,</li> <li>Longitudinale,</li> <li>Monocentrique,</li> <li>A visée fondamentale.</li> </ul> </li> <li>Tous les patients inclus dans cette recherche devront vérifier tous les critères d'inclusion listés ci-dessous : <ul> <li>Consentement écrit donné par le participant,</li> <li>Patient de 18 ans et plus,</li> </ul> </li> </ol> |
| SCHEMA DE L'ETUDE CLINIQUE | <ol> <li>Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation avec la persistance des LT CART-BCMA (mesurée par le pourcentage de LT CAR-BCMA(+)) dans la moelle osseuse à M3 et à M12.</li> <li>Mesure des concentrations de cytokines (sCD95L, IL-1β, IFN-γ, IL-6, IL-10, IL-15 et TNF-α) dans le sérum des patients avant aphérèse et à chaque temps après injection du produit CART-BCMA et corrélation avec le pourcentage de LT CAR-BCMA(+) des LT CAR-BCMA(+) en périphérie et/ou dans la moelle osseuse.</li> <li>Il s'agit d'une étude prospective interventionnelle avec risques et contraintes minimes de catégorie 2, descriptive Exploratoire, <ul> <li>Non randomisée,</li> <li>Longitudinale,</li> <li>Monocentrique,</li> <li>A visée fondamentale.</li> </ul> </li> <li>Tous les patients inclus dans cette recherche devront vérifier tous les critères d'inclusion listés ci-dessous : <ul> <li>Consentement écrit donné par le participant,</li> </ul> </li> </ol> |





| | <ul> <li>4) Patient allant recevoir un CAR-T en suivant les règles et autorisations en vigueur en France.</li> <li>5) Patient bénéficiant de la sécurité sociale</li> </ul> |
|---|---|
| CRITERES DE NON INCLUSION | <ul> <li>Tous les patients inclus dans cette recherche ne devront avoir aucun des critères de non inclusion listés ci-dessous :</li> <li>1) Patient ayant une santé physique et/ou psychologique sévèrement altérée, qui selon, l'investigateur, peut affecter la compliance du participant à l'étude.</li> <li>2) Participation simultanément à une autre étude comprenant une période d'exclusion toujours en cours</li> <li>3) Personne bénéficiant d'une protection renforcée à savoir les mineurs, les femmes enceintes et/ou allaitantes, les personnes privées de liberté par une décision judiciaire ou administrative, les personnes séjournant dans un établissement sanitaire ou social, les majeurs sous protection légale et enfin les malades en situation d'urgence;</li> </ul> |
| TAILLE D'ETUDE | 60 patients inclus pour obtenir 40 patients analysables au final. |
| DUREE DE L'ETUDE CLINIQUE | Durée de la période d'inclusion : 48 mois Durée de participation de chaque participant : maximum 27 mois |



CART-I5M

| Γ | |
|---|---|
| | Durée totale de l'étude clinique : 87 mois au total (soit 48 mois d'inclusion, 27 mois de suivi et 12 mois d'analyses). |
| ANALYSE STATISTIQUE DES DONNEES | Il s'agit d'une étude à visée fondamentale. Les analyses seront menées sous GraphPad PrismV8.2.1 (GraphPad Software, San Diego California, USA) et SASv9.4 (NYC, CAL). Utilisation des méthodes descriptives usuelles (moyenne, écart type, fréquence). Les comparaisons de moyennes seront réalisées par un t test de de Student et les comparaisons de fréquence par la méthode du chi² d'indépendance. Les données non normalement distribuées seront analysées par un test de Mann-Whitney U pour les variables quantitatives. Les études de corrélations seront évaluées par les coefficients de corrélation de Spearman pour les variables quantitatives. Toutes les analyses seront réalisées avec un risque alpha bilatéral de 0,05. Il n'y aura pas d'analyses intermédiaires. |
| RETOMBEES ATTENDUES | Notre programme de recherche devrait contribuer à optimiser l'efficacité du traitement par les cellules CAR-T, ceci en identifiant les éléments cellulaires associés au succès et à la pérennité du traitement par les LT CAR-BCMA. D'un point de vue biologique, nous présumons que la longévité/survie des cellules CAR-T sera étroitement associée au statut souche (ou stemness) initial des lymphocytes utilisés lors de l'aphérèse. Dans l'affirmative, les résultats obtenus devraient permettre de mieux orienter lors de leur production la composition des cellules CAR-T infusées; en effet, nous présumons que la nature des LT du patient qui sont récupérés, modifiés génétiquement en culture, multipliés puis réinjectés chez le patient, contribue significativement à l'hétérogénéité des réponses cliniques. In fine, nous attendons que l'acquisition de fonctions effectrices et/ou le maintien d'un état souche au sein des cellules CAR-T(+) et/ou des cellules CART(-) via des effets bystanders, sera(seront) corrélé(s) à une meilleure réponse complète clinique et durable. A côté de leur caractère translationnel, nos travaux d'immunobiologie pourraient avoir un aspect novateur et cognitif en contribuant à une meilleure connaissance des éléments cellulaires LTI et des mécanismes sous-jacents mis en jeu dans le contrôle du MM. En retour, nous postulons que notre étude longitudinale des CAR-T et de leur signature associée au maintien d'une réponse clinique et durable, contribuera au développement de futures thérapies ciblées, y compris de cellules CAR-T de nouvelle génération |





# 2 JUSTIFICATION SCIENTIFIQUE ET DESCRIPTION GENERALE

# 2.1 Etat actuel des connaissances

# 2.1.1 Sur la pathologie

Le myélome multiple (MM) est une hémopathie maligne chronique, définie par la prolifération monoclonale dans la moelle osseuse (MO), de plasmocytes transformés (PCs)qui sécrètent une immunoglobuline monoclonale (Igmo), complète ou, plus rarement, incomplète (myélome à chaînes légères, 30% des cas).

Le MM représente la deuxième hémopathie maligne la plus fréquente après les lymphomes, soit 10% des hémopathies malignes et 1% des cancers (Siegel et al. 2019) et est responsable de 4,1 décès pour 100 000 habitants chaque année (Moreau et al. 2017).

La gammapathie monoclonale de signification indéterminée (GMSI ou MGUS en anglais) précède toujours l'apparition d'un myélome, même si son diagnostic passe parfois inaperçu. Découverte le plus souvent fortuitement à l'occasion d'un examen sanguin, cette anomalie bénigne n'entraîne pas de symptôme : il s'agit de la présence d'un clone de plasmocytes dans la moelle osseuse en quantité anormale.

Elle concerne plus de 3 % des personnes âgées de plus de cinquante ans. Sur l'ensemble des patients concernés, seule une petite proportion verra leur GMSI évoluer en myélome et aucun signe ne permet d'identifier les profils à risque. Dans la grande majorité des cas de myélome, on ne retrouve pas d'antécédents familiaux.

Les manifestations clinico-biologiques liées au MM résultent de différents facteurs, notamment l'excès d'Igmo sécrétée (insuffisance rénale, hyperviscosité, etc), l'infiltration de la moelle osseuse par les PCs (anémie, atteinte osseuse) et la sécrétion de différentes cytokines par ces dernières. Au-delà du pronostic initial de la maladie, un facteur pronostic déterminant est la réponse au traitement (pour revue, (Kumar et al. 2017)) dont la profondeur est corrélée à la survie.

Malgré d'important progrès thérapeutiques au cours des dernières années, le MM reste incurable et les rechutes, parfois plusieurs années après la fin du traitement, sont inévitables. La prolifération des PCs se déroule au sein d'un micro-environnement médullaire (MEM) osseux, mettant en jeu des interactions avec des cellules du stroma médullaire, des cellules immunitaires, y compris des lymphocytes. Ces interactions dépendent de l'action de très nombreuses cytokines et chémokines agissant sur les PCs et sur les différents partenaires cellulaires du MEM, notamment les lymphocytes T et les NK.

### 2.1.2 <u>L'immuno-vigilance et immuno-édition : application au myélome multiple</u>

Le développement d'une tumeur suit trois étapes successives qui s'intègrent dans la théorie dite des « 3 E » : Équilibre, Edition, Échappement (Dunn et al. 2004). Cette théorie illustre les interactions entre le système immunitaire et le cancer au cours de la genèse de ce dernier.

Le MM est un bon exemple d'application de cette théorie des « 3 E » car il s'inscrit dans un groupe de maladies dénommées « gammapathies monoclonales » avec un *continuum* entre le stade MGUS ou gammapathie de signification indéterminée, le sMM ou MM indolent et le MM symptomatique (Kumar et al. 2017; Rajkumar 2016).

En effet, au stade MGUS, le clone plasmocytaire existe avec une production d'Ig monoclonale complète ou non, dosable dans le sang périphérique mais la prolifération des plasmocytes au niveau médullaire est contrôlée par le système immunitaire. Ce stade correspond à la phase d'Élimination. Le stade MGUS est

Version n°2 du 08.10.2025 CONFIDENTIEL Page 12 sur 54





considéré comme un état pré-cancéreux qui précède systématiquement l'apparition du MM avec un risque d'évolution vers le MM d'environ 1% par an. En cas d'évolution vers le sMM, le clone devient tumoral avec la présence de 10% de plasmocytes de la MO mais il persiste une forme d'immuno-surveillance dont le caractère asymptomatique du sMM est le témoin. Ce stade correspond à la phase d'*Équilibre*.

Enfin la progression vers le stade du MM symptomatique cliniquement correspond à la phase d'*Échappement*. A ce stade, les plasmocytes malins sont devenus immuno-résistants et échappent au système immunitaire, voire sont capables de contourner celui-ci. En outre, le plasmocyte malin *via* la production de cytokines, va modifier les caractéristiques du MEM pour favoriser sa survie et sa prolifération. Ces modifications vont également être impliquées dans le développement de mécanismes de résistance aux différentes drogues auxquelles le MM va être exposé au cours de la prise en charge.

Bien que les mécanismes cellulaires de l'immuno-surveillance dans le MM ne soient pas totalement élucidés, l'apparition de la maladie semble en partie dépendre de la perte de fonctions des LT CD8 résidents médullaires (Chang et al. 2018) tandis que le rôle des lymphocytes T innés dans l'immunité anti-myélome a déjà été démontrée (Favreau et al. 2017).

# Les principaux marqueurs des plasmocytes tumoraux :

Le Pc, cellule tumorale du MM, est caractérisée sur le plan cytologique par son caractère dystrophique et par l'expression des marqueurs CD38 et CD138.

Le premier, CD38, est une ectoenzyme impliquée dans la synthèse d'ADP-ribose dont l'expression est beaucoup plus élevée à la surface des Pc qu'à la surface des plasmocytes sains ce qui en fait une cible thérapeutique pour le Daratumumab (un anticorps monoclonal thérapeutique) (Kumar et al. 2017; Rajkumar 2016).

Le second, CD138, appartient à la famille des syndecans qui sont impliquées dans la prolifération, la migration et l'interaction avec la matrice extracellulaire.

Un autre marqueur d'intérêt est BCMA (pour B-cell maturation antigen), une molécule appartenant à la superfamille des récepteurs du TNF, exprimée par différentes sous-populations de lymphocytes B différenciés et par les Pc malins au cours du MM. BCMA transduit des signaux de survie pour les Pc du MM par l'interaction avec ses ligands BAFF (pour B-cell activating factor) et APRIL (pour a proliferation inducing ligand). BCMA peut être l'objet d'un shedding aboutissant à la production d'une forme soluble de BCMA (sBCMA) qui est un reflet de la masse tumorale du MM et un potentiel élément d'interférence avec les traitements ciblant BCMA.

### Traitement du MM:

Selon les recommandations de l'IMWG (*International myeloma working group*) (Rajkumar 2016), le diagnostic de MM nécessite la réalisation d'un myélogramme qui retrouve la présence d'au moins 10% de plasmocytes dans la MO.

Les manifestations clinico-biologiques, sont l'hyperCalcémie, l'insuffisance Rénale, l'Anémie et les lésions ostéolytiques (*Bone lesions*) (critères dits *CRAB*). Lorsque l'un de ces symptômes est présent, le MM est alors dit « symptomatique » et requiert un traitement (Rajkumar 2016).

Ces critères de traitement historiques ont été plus récemment complétés par les critères *SLIM CRAB* qui comprennent un *ratio* des chaînes légères > 100, une plasmocytose médullaire clonale supérieure à 60% et une image nodulaire focale à l'IRM médullaire.

L'adjonction de ces critères *SLIM CRAB*, qui sont le reflet d'une maladie biologiquement active, ont donc l'avantage de permettre l'initiation plus précoce d'un traitement et ce avant l'apparition de lésions d'organe.

Version n°2 du 08.10.2025 CONFIDENTIEL Page 13 sur 54





En l'absence de critères *SLIM CRAB*, le MM est défini comme « indolent » (sMM, *smoldering multiple myeloma*) (Rajkumar 2016). Actuellement, les patients au stade de sMM, en dehors d'essais thérapeutiques, requièrent seulement une surveillance, sans la mise en place d'un traitement, même si ce concept devrait rapidement évoluer, pour certains patients avec un sMM de haut risque évolutif (cf ASH 2024 essai AQUILA phase 3) (Rajkumar 2016).

Le traitement du MM en première ligne repose aujourd'hui principalement sur des thérapies ciblées (inhibiteurs du protéasome, immunomodulateurs) en association à l'immunothérapie avec les anticorps monoclonaux (Mab) anti-CD38 (Dimopoulos et al. 2021).

Selon l'âge (généralement <65-70 ans) et l'état général, une autogreffe de cellules souches hématopoïétiques après une chimiothérapie intensive myéloablative par *Melphalan* haute dose peut être proposée.

L'autogreffe intervient après une phase de traitement d'induction (4-6 cycles) reposant sur l'association thérapies ciblées et immunothérapie. Après l'autogreffe les patients reçoivent un traitement de maintenance pour 2 à 3 ans. Chez les patients plus âgés (non éligibles à l'autogreffe), on propose un traitement de 3 à 4 molécules (association d'immunothérapie et thérapies ciblées) en continu, c'est-à-dire jusqu'à progression.

A la rechute, les immunothérapies de « nouvelle génération » s'imposent avec :

- Les Ac bispécifiques comme le Teclistamab, résultent de la fusion de 2 MAb connectés entre eux par un peptide. Par leur structure coudée et leur capacité à cibler simultanément le CD3 des LT et un Ag à la surface de la cellule cible (le BCMA, un récepteur du TNF exprimé préférentiellement dans les LB matures dont les plasmocytes malins), ils permettent de rapprocher les LT cytotoxiques de la cellule tumorale et d'induire leur activation et provoquer la lyse des plasmocytes myélomateux.
- Les cellules CAR-T comme l'*Idecabtagene vicleucel* ou Ide-cel (Munshi et al. 2020) et le *ciltacabtagene autoleucel* ou cilta-cel qui sont des LT autologues collectés par aphérèse et, qui après modification génétique, expriment un récepteur chimérique portant des domaines variables d'un mAb dirigé contre BCMA à la surface des plasmocytes malins et des domaines de transduction qui induisent l'activation des cellules CART et la lyse des cellules tumorales.

Ces innovations thérapeutiques, en mettant en jeu les LT présents au sein de la niche médullaire, montrent l'importance de connaitre au mieux la physiologie et les mécanismes d'action du SI dans le MM. Car le but de ces immunothérapies est de restaurer l'efficacité du système immunitaire contre le cancer et de repousser au maximum la rechute voir de viser la rémission définitive par le contrôle pérenne de la tumeur résiduelle.

# 2.1.3 Sur la stratégie et/ou les procédures de référence à l'étude

### La place des cellules CAR-T dans la thérapeutique du MM:

Depuis l'émergence de l'immunothérapie et notamment des Ac monoclonaux anti-CD38 la survie des patients s'est nettement allongée. Cependant, tous les patients sont à risque de rechute, la plupart présenteront même plusieurs rechutes au cours de l'histoire de leur maladie.

Les stratégies à la rechute doivent donc être nombreuses et potentiellement cibler des antigènes ou des mécanismes différents des molécules utilisées dans les premières lignes.

A ce titre, ces dernières années ont été marqué par l'apparition de nouvelles classes thérapeutiques comme : les anticorps conjugués (ou ADC pour antibody drug conjugate) qui permettent de coupler une molécule cytotoxique à un anticorps (Ac), les Ac bispécifiques qui permettent de rapprocher via le CD3 les lymphocytes T (LT) de la cellule tumorale, d'induire l'activation des LT et de provoquer la lyse des cellules tumorales, ou encore les CAR-T cells. Les cellules CART (pour Chimeric Antigen Receptor) : sont

Version n°2 du 08.10.2025 CONFIDENTIEL Page 14 sur 54





développés à partir de LT autologues collectés par lymphaphérèse et génétiquement modifiés pour exprimer un CAR, autrement dit un récepteur synthétique chimérique qui porte les domaines variables de chaînes légères et lourdes d'un anticorps monoclonal spécifique d'un antigène tumoral, les domaines de transductions de CD3z (CD247) et de costimulation de CD28 ou de CD137 (4.1.BB).

Les domaines variables permettent la reconnaissance de l'antigène à la surface des cellules tumorales tandis que les domaines de transduction et de costimulation induisent l'activation des cellules CART, leur prolifération et la lyse des cellules tumorales (pour revue, (Majzner and Mackall 2019)).

Les cellules CART anti-CD19 (CAR-CD19) utilisés dans le traitement des syndrome lymphoprolifératifs B ont été les premiers pour lesquels une efficacité clinique incontestable ait été décrite (pour revue, (Majzner and Mackall 2019; Brown and Mackall 2019)).

Cependant, dans bon nombre de cas, les rémissions obtenues sont transitoires et il a été observé un épuisement des cellules CART anti-CD19 chez les patients qui ne répondent pas au traitement (pour revue, (Majzner and Mackall 2019)). Ainsi, les taux de réponse et la survie des patients, au-delà des caractéristiques de la pathologie sous-jacente et du produit CART utilisé, semblent corrélés à la persistance des cellules CAR T suggérant la mise en place de mécanismes d'homéostasie particuliers à chaque patient.

# <u>Le statut immunitaire initial du patient et la signature mémoire portée par les cellules CART comme éléments déterminant leur longévité et efficacité ?</u>

Des travaux récents en modélisation animale soulignent que l'épuisement des cellules CAR-T est associé/dû à une exhaustion phénotypique et métabolique (Abken 2016; Kawalekar et al. 2016). Fait remarquable, les cellules LT CAR-CD19 associées aux rémissions les plus longues étaient celles qui avaient un phénotype de type centrale-mémoire (CM), conservant une plus grande plasticité et un plus large potentiel de différenciation grâce à un contingent souche de cellules TSCM (Stem Cell Memory) que celles qui avaient un phénotype de type mémoire-effecteur (ME) ou mémoire en différenciation terminale (Abken 2016; Kawalekar et al. 2016), l'équivalent des cellules EMRA (effector-memory exprimant CD45RA) décrites au sein des LT CD8 humains.

Ces TSCM ont les caractéristiques des cellules T naïves (TN : CD45RA+CCR7+CD62L+CD28+) associées à des quantités significatives de CD122 (IL-2Rb) et de CD95 avec des propriétés de renouvellement et une forte capacité d'expansion (Gattinoni et al. 2011). En parallèle, certaines cellules T non conventionnelles, à cheval entre l'immunité innée (cellules NK) et l'immunité adaptative (cellules T CD4+ et CD8+) exercent des fonctions antitumorales. Il s'agit notamment des cellules NKT et T CD8+ innées, des cellules T invariantes associées aux muqueuses (MAIT), et des cellules T-γδ.

De plus, dans les mêmes travaux, il existait une meilleure efficacité métabolique et un meilleur maintien des LT CAR-CD19 CM quand le récepteur chimérique utilisait le domaine de costimulation de CD137 plutôt que celui de CD28. Plus récemment, l'équipe de Carl June (Good et al. 2021) a apporté des arguments suggérant que l'acquisition d'un phénotype EMRA par les LT CAR-CD19 et leur épuisement étaient corrélés à l'expression de marqueurs NK.

Cette transition phénotypique des LT CAR-CD19 d'un phénotype « T CD8-like » vers un phénotype « NK-like » était observée tant dans un modèle *in vitro* de CART humains dirigés contre un antigène de mésothéliome que *in vivo* chez des patients traités par des LT autologues CAR-CD19 utilisant le domaine de costimulation de CD137 (CAR-CD19 tisagenlecleucel). L'hypothèse proposée par les auteurs était que la stimulation chronique des cellules CAR-T était responsable de cette transition d'un statut « adaptatif » T-CD8 vers un statut « inné »-NK-like.

Une autre théorie serait celle de la « precocious differentiation » proposée par les travaux de Restifo et Klebanoff en thérapie cellulaire adoptive (Klebanoff et al. 2016) et par cellules CART (Yi et al. 2024) chez

Version n°2 du 08.10.2025 CONFIDENTIEL Page 15 sur 54





la souris. Le couple CD95, CD95 ligand (CD95L) pourrait jouer un rôle majeur dans la persistance des cellules CAR T via une voie moléculaire qui reste à définir. En effet, il a été montré in vitro et dans des modèles murins que l'expression de CD95L peut accélérer, par contact cellulaire, la différenciation des cellules CAR T (en TEM/TEMRA) et interrompre la réponse immunitaire, compromettant la réponse antitumorale.

Les caractéristiques des lymphocytes sont donc susceptibles d'intervenir dans la qualité du CAR-T qui sera produit. A cet égard, le travail de Chen et al. 2021 (Chen et al. 2021) suggère que le succès du traitement par les CAR-CD19 chez l'humain est associé au maintien de l'expression du facteur de transcription TCF1 (dont le gène est *Tcf7*) parmi les cellules utilisées pour la fabrication des cellules thérapeutiques. Or ce facteur est justement impliqué dans le maintien des lymphocytes naïfs et CM. Par ailleurs, chez deux patients traités par CAR-CD19 et ayant une rémission supérieure à 10 ans, des cellules chimériques à des fréquences d'environ 1-1,5% sont observables dans le sang et correspondent à des cellules CAR-CD19(+) CD4(+) et/ou TCR-γδ.

De façon intéressante, ces cellules CAR-CD19(+) CD4(+) chez ces deux patients ont un phénotype de cellules cytotoxiques (Melenhorst et al. 2022). Ces résultats renforcent l'hypothèse que la qualité des cellules transduites par le récepteur chimérique joue un rôle déterminant et qu'il est essentiel d'évaluer l'état du système immunitaire avant d'initier un traitement par cellules CART.

L'ensemble de ces données conduit à proposer que l'efficacité des cellules CART pourrait reposer sur l'existence d'un pool initial ayant un potentiel de *stemness*, en équilibre subtil entre un statut de maintien par prolifération et un flux basal et continu de différenciation en cellules effectrices. Un pool initial de cellules CAR-T avec un potentiel de *stemness* altéré favoriserait alors l'accumulation de cellules CART effectrices en exhaustion et leur disparition. L'expression plus importante de CD95L à la surface des lymphocytes T (CAR et non CAR) pourrait également favoriser la différenciation précoce des cellules effectrices.

### **Modes d'action des cellules CAR-T:**

Il est bien reconnu que les CART peuvent agir par une cytotoxicité directe sur les cellules tumorales (pour revue, (Majzner and Mackall 2019; Cazaux et al. 2019)).

Cependant, des travaux récents redéfinissent le mode d'action des cellules CART en montrant aussi leur capacité à recruter des LT non chimériques, procédant ainsi à une sorte de « reset » de la réponse immunitaire.

A cet égard, on retiendra en particulier la démonstration récente chez l'humain que la rémission associée au traitement d'un glioblastome par un CAR anti-IL-13Ra2 est retrouvée corrélée à une intense réponse des LT CAR(-) et à une activation de cellules myéloïdes anti-tumorales.

Cette activation bystander des LT et des cellules myéloïdes dépend de l'IFN- $\gamma$  des cellules CART(+) (Alizadeh et al. 2021).

Ainsi, les cellules CAR-T dialoguent étroitement avec l'environnement immunitaire, y compris via la production de cytokines, et ce dialogue est essentiel pour leur activité thérapeutique.

# <u>Caractéristiques des CART (LT CAR-BCMA) utilisés dans le traitement du MM :</u>

Différents antigènes tumoraux de PCs de MM ont été envisagées comme cibles de cellules CART, parmi ceux-ci, le BCMA est l'antigène pour lequel s'est mis en place un consensus, la plupart des CART développés dans le traitement du MM sont dirigés contre cet antigène; nous les noterons CAR-BCMA. Le service d'hématologie et thérapie cellulaire du CHU de Poitiers participe à deux études de phase 3 internationales utilisant la technologie CART anti-BCMA: l'étude CARTITUDE-5 (pour « A Study of Bortezomib, Lenalidomide and Dexamethasone (VRd) Followed by Cilta-cel, a CAR-T Therapy Directed Against BCMA Versus VRd Followed by Lenalidomide and Dexamethasone (Rd) Therapy in Participants With Newly Diagnosed Multiple Myeloma for Whom ASCT is Not Planned as Initial Therapy ») et l'étude KarMMa-9 (« A Study to Compare the Efficacy and Safety of Idecabtagene Vicleucel With Lenalidomide

Version n°2 du 08.10.2025 CONFIDENTIEL Page **16** sur **54** 





Maintenance Therapy Versus Lenalidomide Maintenance Therapy Alone in Adult Participants With Newly Diagnosed Multiple Myeloma Who Have Suboptimal Response After Autologous Stem Cell Transplantation"). Nous allons brièvement décrire les caractéristiques de ces CAR T et le but de ces études cliniques.

# 1) L'étude CARTITUDE-5 et le Ciltacbtagene (Cilta-cel ou autoleucel).

Le but de cette étude est de comparer l'efficacité de l'induction du bortezomib, du lenalidomide et de la dexaméthasone (VRd) suivie d'une administration unique de ciltacabtagene autoleucel (cilta-cel) versus induction du VRd suivie d'un entretien par lenalidomide et dexaméthasone (Rd) dans le MM nouvellement diagnostiqué chez des patients pour lesquels l'allotransplantation de cellules souches (ASCT) n'est pas prévue comme traitement initial en termes de survie sans progression (SSP).

Ce CAR utilise deux domaines variables VHH de lama en tandem spécifiques de deux épitopes différents de BCMA. Cette particularité confère au Cilta-cel une affinité potentielle plus élevée pour l'antigène cible. Ce CAR utilise de façon classique le domaine intracellulaire CD247 permettant la transduction du signal lors de l'engagement du CAR et le domaine de costimulation de CD137 (pour revue, (Manier et al. 2022)).

Après 8 cycles de VRd, le conditionnement/la lymphodéplétion précédant l'injection des cellules thérapeutiques utilise une combinaison Fludarabine et de Cyclophospamide, 0,75.106cellules CART positives/kg sont ensuite injectées au patient. Les patients du bras contrôle, après les 8 cycles de VRd, reçoivent comme traitement d'entretien du Lenalidomide avec de la dexaméthasone (Rd).

# 2) L'étude KarMMa-9 et l'IdecCabtagene (Ide-cel)).

Cet essai clinique randomisé de phase 3 utilise un CAR dont le récepteur chimérique est formé des domaines variables de chaînes lourdes et de chaînes légères d'un Ac murin spécifique d'un épitope de BCMA; Les unités de transduction et de costimulation sont similaires à celles du Cilta-cel.

Le conditionnement/la lymphodéplétion précédant l'injection des cellules thérapeutiques utilise une combinaison Fludarabine, Cyclophospamide (jour (J)-5, J-4, J-3). Au J0 du traitement, selon la masse corporelle du patient, 150 à 450. 106 cellules chimériques sont injectées, les cellules CAR-BCMA(+) représentant 60 à 70 % des cellules injectées. Le pic d'expansion des cellules chimériques est observé vers J10/J11.

Le conditionnement suit les mêmes principes que pour l'Ide-cel, la principale différence étant le nombre de cellules CAR-Tl injectées à J0, réduite à 50 à 70. 106 cellules transduites par le CAR-BCMA selon la masse corporelle du patient.

L'efficacité thérapeutique des deux CAR-BCMA est remarquable avec un ORR de 80% avec l'ide-cel et de 90% avec le cilta-cel. Plusieurs arguments suggèrent que le Cilta-cel a un potentiel d'expansion *in vivo* plus important que l'Idecel (pour revue, (Manier et al. 2022)).

Les taux de réponse et la survie des patients, au-delà des caractéristiques du MM, semblent corrélés à la capacité d'expansion, à la persistance et à la fonctionnalité des cellules CAR-T.

# 2.2 Hypothèse de l'étude clinique et résultats attendus

Nous émettons ici l'hypothèse principale que le caractère souche (ou *stemness*) des LT avant l'aphérèse et son maintien après activation/stimulation peut prédire la persistance des LT CAR-BCMA chez le patient, un critère reconnu de la bonne réponse au traitement par cette thérapie.

Version n°2 du 08.10.2025 CONFIDENTIEL Page 17 sur 54





Dans le cadre du présent projet, nous testerons cinq mécanismes non exclusifs susceptibles d'être impliqués dans la réussite du traitement :

- 1) le maintien d'une signature CM TCF1(+) dans les LT utilisés pour la fabrication des LT CAR-BCMA qui serait associé à une meilleure efficacité du CAR chez le patient (maintien en nombre, en fonctions effectrices et en potentiel prolifératif/survie);
- 2) le maintien des fonctions effectrices et de l'expansion des LT CAR-BCMA après leur administration aux patients qui serait contrôlé par une balance entre le maintien de l'expression de TCF1 et de celle des facteurs de transcription (Eomes, T-bet, Helios) associés à l'acquisition de fonctions effectrices et cytotoxiques (perforine, granzymes, expression de l'IFN-g et du TNF-α)
- 3) le recrutement bystander de LT CAR-T(-) anti-tumoraux qui serait contrôlé par les LT CAR-BCMA(+).
- 4) l'expression de CD95L membranaire et la différenciation précoce (precocious differentiation), qui pourrait interférer avec la persistance des LT CAR-BCMA(+) dans le sang périphérique aux différents temps du suivi longitudinal sur 1 an
- 5) le profil inflammatoire des patients, déterminé par dosages cytokiniques (sCD95L, IL-1 $\beta$ , IFN- $\gamma$ , IL-6, IL-10, IL-15 et TNF- $\alpha$ ) à chaque temps et sa corrélation avec la persistance des LT CAR-BCMA(+) en périphérie et/ou dans la moelle osseuse.

# 2.3 Bénéfices / risque

#### 2.3.1 Bénéfices

# 2.3.1.1 Bénéfices attendus pour le patient

Il n'y a pas de bénéfice individuel direct pour les patients.

### 2.3.1.2 Bénéfices attendus pour la société

Les retombées socio-économiques attendues sont :

- de proposer un/des nouveaux marqueurs cellulaires prédictifs permettant de guider le choix des traitements dans le MM (dépôt de brevet possible).

### 2.3.1.3 Bénéfices attendus pour la communauté médicale

Le projet proposé pourra contribuer à une meilleure prise en charge des patients en termes de soins dans le domaine de l'oncologie, ceci en identifiant des marqueurs cellulaires immunologique prédictifs d'une réponse efficace aux traitements anti cancéreux et/ou à un ciblage immuno-thérapeutique.

#### 2.3.2 Risques

Les risques encourus par les patients pour la recherche sont minimes puisque nous nous adosserons à des prélèvements déjà réalisés dans le soin courant.

# Recueil de sang supplémentaire :

On peut observer un hématome au point de ponction, une légère douleur, un léger saignement, voir un malaise.

# Recueil de ponction de moelle osseuse supplémentaire :

Les complications liées à ce geste sont très rares et sont les suivantes :

- Saignement local : un pansement compressif peut être nécessaire,
- Douleur résiduelle : cède en général aux analgésiques de type paracétamol,

Version n°2 du 08.10.2025 CONFIDENTIEL Page 18 sur 54





- Infection : pour l'éviter, il faut respecter des conditions strictes d'asepsie,
- Disjonction manubrio-corporéale : en cas de fragilité osseuse,
- Tamponnade par hémopéricarde : rarement décrite lors des prélèvements au niveau du manubrium,
- Pneumopéricarde,
- Pneumothorax,
- Rupture du trocar.

L'investigateur doit constamment surveiller, évaluer et documenter les risques et doit s'assurer qu'ils pourront être gérés de manière satisfaisante.

# 2.4 Retombées attendues

Malgré une nette amélioration de la survie des patients atteints de myélome multiple en rechute grâce à la thérapie par CAR T cells, l'optimisation de leur activité antitumorale reste un enjeu de premier plan.

Sur le plan fondamental, le projet devrait ouvrir de nouvelles perspectives pour une meilleure compréhension :

- des mécanismes immunitaires contrôlant les tumeurs ainsi que des modes d'action des immunothérapies anti-cancéreuses utilisant la thérapie cellulaire par CAR-T,
- des modes d'activation et d'exhaustion des LTI au cours des processus tumoraux.

Les retombées socio-économiques attendues sont :

- de proposer un/des nouveaux marqueurs cellulaires prédictifs permettant de guider le choix des traitements dans le MM (dépôt de brevet possible).

# 2.5 <u>Justification du faible niveau d'intervention</u>

Les patients font l'objet de prélèvements biologiques et d'une consultation permettant la prise en charge thérapeutique par cellules CART anti-BCMA dans le Myélome Multiple dans le cadre du soin courant. Pour répondre aux objectifs de l'étude, il sera effectué, aux patients en plus de leur bilan biologique classique, un recueil de sang périphérique afin d'effectuer les analyses prévues. Ces recueils de sang supplémentaires devront être effectués au maximum lors de prises de sang de soin courant. Dans de rares cas, un recueil spécifique pour l'étude pourrait avoir lieu.

Aucune administration de substances ne sera effectuée et la prise en charge du patient ne sera pas modifiée.

Une ponction de moelle osseuse est prévue dans les soins courants du suivi du traitement par thérapie CART anti-BCMA. Lors de ce prélèvement, 3 à 5 ml supplémentaires seront recueillis.

Le recueil supplémentaire de moelle osseuse réalisé pour répondre aux objectifs de l'étude lors d'un prélèvement requis dans le cadre du soin et la possibilité d'un recueil spécifique de sang hors bilan de soin courant, font que le projet entre dans les actes listés dans l'arrêté du 12 avril 2018, fixant la liste des recherches mentionnées au 2° de l'article L1121-1 du code de la santé publique :

- Les prélèvements de sang effectués spécifiquement pour la recherche qui sont réalisés par ponction veineuse, périphérique ou capillaire
- Les prélèvements d'échantillons biologiques, autres que le sang, spécifiquement pour les besoins de la recherche :

Version n°2 du 08.10.2025 CONFIDENTIEL Page 19 sur 54





\*tissus ou biopsies élargis ou supplémentaires à l'occasion de gestes médico-chirurgicaux réalisés dans le cadre du soin

Ce protocole s'inscrit donc dans une recherche à risques et contraintes minimes (RIPH2).

Version n°2 du 08.10.2025 CONFIDENTIEL Page **20** sur **54** 





# 3 OBJECTIFS ET CRITERE DE JUGEMENT PRINCIPAL

# 3.1 Objectif principal

Sur notre cohorte de patient atteint d'un MM et traités par thérapie CART-BCMA, notre objectif principal est de pouvoir corréler le caractère souche (ou *stemness*), reflété par l'expression du facteur de transcription TCF1, des lymphocytes T (CD3+) avant l'aphérèse destinée à la production du CAR-BCMA, avec : 1) la persistance des lymphocytes CAR-BCMA chez le patient, dans le sang périphérique aux différents temps du suivi longitudinal sur 1 an (J10, M1, M3, M6 et M12) ; 2) la réponse à la thérapie CAR-T anti-BCMA.

# 3.2 Critère de jugement principal :

- 1) Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation avec le pourcentage de LT CAR-BCMA(+) aux différents temps de suivi sur un an.
- 2) Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation avec la réussite du traitement, définie par une rémission du MM, telles que définies par les recommandations internationales (IMWG).

Les critères biologiques seront obtenus par des expériences de cytométrie en flux, qui seront conduites au laboratoire INSERM U1313, et sur la plateforme d'Imagerie de l'Université de Poitiers, ImageUP, sur le cytomètre spectral Aurora (Cytek).

L'équipe utilise des protocoles de marquage standardisés des cellules immunitaires, avec des marqueurs reconnus et un suivi des lots d'anticorps utilisés.

Le cytomètre spectral de la plateforme ImageUP est calibré à chaque utilisation selon les recommandations du fabriquant et une maintenance bisannuelle est effectuée. Pour limiter la variabilité inter-expérience, toutes les manipulations seront confiées à un/une technicien(ne) de recherche formée au laboratoire INSERM U1313, recruté spécifiquement pour ce projet.

#### Critères cliniques selon le groupe international du MM (IMWG) :

Rémission complète (CR) : Immunofixation négative sur le sérum et l'urine et disparition de tout plasmacytome des tissus mous et moins de 5% de cellules plasmatiques dans la moelle osseuse (Kumar etal., 2016).

Version n°2 du 08.10.2025 CONFIDENTIEL Page **21** sur **54** 





# 4 OBJECTIFS ET CRITERES DE JUGEMENT SECONDAIRES

# 4.1 **Objectifs secondaires**

- 1. Déterminer si le caractère souche ou *stemness*, reflété par l'expression du facteur de transcription TCF1, des lymphocytes T (CD3+) avant l'aphérèse et/ou la lymphodéplétion, est corrélé avec la persistance des lymphocytes CAR-BCMA chez le patient, dans la moelle osseuse à M3 et à M12.
- 2. Identifier les mécanismes d'homéostasie de la réponse immunitaire, reflétés par l'expression de CD95L membranaire et la différenciation précoce (precocious differentiation), interférent avec la persistance des LT CAR-BCMA(+) dans le sang périphérique aux différents temps du suivi longitudinal sur 1 an ;
- 3. Déterminer si le profil inflammatoire des patients, déterminé par dosages cytokiniques (sCD95L, IL-1β, IFN-γ, IL-6, IL-10, IL-15 et TNF-α) à chaque temps est corrélé avec la persistance des LT CAR-BCMA(+) en périphérie et/ou dans la moelle osseuse.

# 4.2 <u>Critères de jugement secondaires</u>

- 1. Analyse longitudinale des pourcentages des LT conventionnels (CD4, Treg, CD8 et leurs différentes sous populations) et non conventionnels (iNKT, LT-γδ, MAIT et LTI CD8) en périphérie et dans la moelle osseuse, dans la fraction CART-BCMA(+) et CART-BCMA(-), de l'expression de CD95 et CD95L membranaire et analyse des fonctions effectrices suivantes :
  - a. État d'exhaustion : expression des marqueurs PD-1, TIM-3, TIGIT, LAG-3
  - b. Arsenal cytotoxique : expression de perforine et de granzymes ;
  - c. Signatures transcriptionnelles: facteurs de transcription Eomes, T-bet, Helios, PLZF.
- 2. Niveau d'expression du facteur de transcription TCF-1 (MFI) dans les lymphocytes T (CD3+) circulant avant l'aphérèse et corrélation avec la persistance des LT CART-BCMA (mesurée par le pourcentage de LT CAR-BCMA(+)) dans la moelle osseuse à M3 et à M12.
- 3. Mesure des concentrations de cytokines (sCD95L, IL-1β, IFN-γ, IL-6, IL-10, IL-15 et TNF-α) dans le sérum des patients avant aphérèse et à chaque temps après injection du produit CART-BCMA et corrélation avec le pourcentage de LT CAR-BCMA en périphérie et/ou dans la moelle osseuse.

Version n°2 du 08.10.2025 CONFIDENTIEL Page 22 sur 54





# 5 CRITERES D'ÉLIGIBILITE

# 5.1 Critères d'inclusion

Tous les patients inclus dans cette recherche devront vérifier tous les critères d'inclusion listés ci-dessous :

- Consentement écrit donné par le participant
- Patient de 18 ans et plus
- Patient ayant un Myélome Multiple selon les recommandations internationales
- Patient allant recevoir un CART BCMA en suivant les règles et autorisations en vigueur en France :
- Patient bénéficiant de la sécurité sociale-

Pour les patients traités par Ide-cel dans le cas de l'accès précoce puis dans la prise en charge dans le droit commun (agrément aux collectivités et prise en charge en sus des GHS) depuis le 12/11/2024 :

ABECMA (idecabtagene vicleucel) est un traitement de 4ème ligne ou plus du myélome multiple en rechute et réfractaire, chez les patients ayant reçu au moins trois traitements antérieurs, incluant un agent immunomodulateur, un inhibiteur de protéasome et un anticorps anti CD38, et dont la maladie a progressé pendant le dernier traitement.

En raison des délais de mise à disposition du produit (comprenant le temps de la détermination de l'éligibilité du patient à un traitement par cellules CAR-T, la leucaphérèse, la production des cellules génétiquement modifiées, la chimiothérapie lymphodéplétive jusqu'à l'acheminement au patient pour la réinjection) et de la toxicité significative à court terme, les patients éligibles à ABECMA (idecabtagene vicleucel) doivent avoir un état général et une espérance de vie compatible avec ces délais.

# 5.2 <u>Critères de non-inclusion</u>

Tous les patients inclus dans cette recherche ne devront avoir aucun des critères de non inclusion listés cidessous:

- Patient ayant une santé physique et/ou psychologique sévèrement altérée, qui selon, l'investigateur, peut affecter la compliance du participant à l'étude.
- Participation simultanément à une autre étude comprenant une période d'exclusion toujours en cours
- Personne bénéficiant d'une protection renforcée à savoir les mineurs, les femmes enceintes et/ou allaitantes, les personnes privées de liberté par une décision judiciaire ou administrative, les personnes séjournant dans un établissement sanitaire ou social, les majeurs sous protection légale et enfin les malades en situation d'urgence ;

# 5.3 <u>Faisabilités et modalités de recrutement</u>

Les patients traités pour un Myélome Multiple sont pris en charge dans le service d'Hématologie, transfusion et Thérapie cellulaire. Actuellement, environ deux patients par mois peuvent bénéficier d'un traitement par CART-BCMA, il est raisonnable d'extrapoler à un recrutement de 10 patients par an, soit 40 patients sur la période de 4 ans d'inclusion de cette étude.

Leurs prises en charge suivent les règles en vigueur en France dans le cadre des plans cancers. La décision thérapeutique relève de la RCP.

Version n°2 du 08.10.2025 CONFIDENTIEL Page 23 sur 54





Le service d'Hématologie, transfusion et Thérapie cellulaire prend en charge les patients de la subdivision Poitou Charentes principalement étant recours pour cette partie de la région NVAQ. Les patients sont identifiés et adressés via la RCP.

La décision thérapeutique de CART suit les recommandations et est proposée aux patients suite à la décision en RCP. Les patients sont ensuite contactés et vu par les équipes médicales et paramédicales selon les recommandation nationales et internationales et en suivant les procédures en vigueur (JACIE).

Lors de ces rencontres avec les patients, en parallèle des différents rendez-vous donnés aux patients pour expliquer les CAR-T, mécanismes, process, étapes, risques, bénéfices, seront évoqués les projets de recherche auxquels le service participe. Il est rappelé au patient qu'il est libre de s'opposer à l'utilisation de son matériel biologique pour la recherche. Un document lui est remis que le patient doit remplir pour se prononcer.

Version n°2 du 08.10.2025 CONFIDENTIEL Page 24 sur 54





# 6 CONCEPTION DE L'ETUDE CLINIQUE

# 6.1 Justification des choix méthodologiques

L'objectif principal étant de comparer les statuts de différentiation, fonctionnels et de stemness des LT CART(+) et CART(-) et de les corréler à la persistance des CART chez le patients, le schéma de l'étude sera transversal, analytique et exploratoire.

Dans le cadre de cette étude, une collection d'échantillons biologiques sera utilisée pour répondre aux différents objectifs de l'étude (Cf. partie 10). Ainsi, environ 25 mL de sang total et 3 à 5 mL de MO seront prélevés à différents temps selon le schéma (cf. partie 6.2) pour tous les sujets inclus dans la présente étude.

Ceci sera nécessaire et suffisant pour extraire les différents éléments biologiques utilisés pour répondre aux objectifs de la présente étude : sérum et cellules mononuclées.

# 6.2 Schéma de l'étude clinique

Il s'agit d'une étude prospective interventionnelle avec risques et contraintes minimes de catégorie 2, descriptive:

- Exploratoire,
- Non randomisée,
- Longitudinale,
- Monocentrique.



Version n°2 du 08.10.2025 CONFIDENTIEL Page 25 sur 54





# 7 DEROULEMENT DE L'ETUDE

# 7.1 <u>Calendrier</u>

Durée de la période d'inclusion : 48 mois

Durée de participation de chaque participant : maximum 27 mois

Durée totale de l'étude clinique : 87 mois au total (soit 48 mois d'inclusion, 27 mois de suivi et 12 mois d'analyses).).





# 7.2 <u>Tableau récapitulatif du suivi participant</u>

| | V0<br>(6 à 8 semaines<br>avant J0) | V1<br>(Environ 1<br>semaine avant<br>J0) | Ј0 | V2<br>(+/- 1j) | V3<br>(+/-5j) | V4<br>(+/- 15j) | V5<br>(+/- 1 mois) | V6<br>(+/- 1<br>mois) | F | U |
|---|---|---|---|---|---|---|---|---|---|---|
| | Inclusion<br>AvAP (*) | AvLD (*) | | J10 | M1 | М3 | M6 | M12 | FU1<br>6 mois | FU2<br>12<br>mois |
| Information/ consentement <sup>(R)</sup> | ✓ | | | | | | | | | |
| Bio collection (R) (Sang périphérique et sérum) | <b>√</b> | ✓ | | ✓ | ✓ | ✓ | <b>√</b> | ✓ | | |
| Bio collection <sup>(R)</sup> (Moelle osseuse) | | ✓ | | | | ✓ | | ✓ | | |
| Histoire de la maladie <sup>(S)</sup> : Diagnostic initial - Date, MGUS, Indolent, plasmocytome isolé, sexe - ISS, R-ISS (β2 microglobuline, albumine, LDH) - Moelle: PM/CMF/risques cytogénétiques sur MO - Sang: Hémoglobine, plaquettes, calcémie, créatinémie, EPS/IFS/FLC - Urines 24h: EPU/IFU - Atteinte osseuse: imagerie (PET/TAP/IRM) + type atteinte, EMD. | <b>V</b> | | | | | | | | | |
| Histoire de la maladie <sup>(S)</sup> : Rechutes - Dates - Moelle: PM/CMF/risques cytogénétiques sur MO - Sang: EPS/IFS/FLC - Urines 24h: EPU/IFU - Traitements | <b>√</b> | | | | | | | | | |
| Thérapie CAR-T cells <sup>(S)</sup> : Diagnostic - Moelle: PM/CMF/risques cytogénétiques sur MO - Sang: EPS/IFS/FLC - Urines 24h: EPU/IFU - Atteinte osseuse: imagerie (PET/TAP/IRM) + type atteinte, EMD | | ✓ | | | | | | | | |
| Thérapie CAR-T cells <sup>(S)</sup> : - Lymphodéplétion - Traitement d'attente - Injection CAR-T (S) | | <b>√</b> | | | | | | | | |
| Evaluation de la réponse suivant IMGW(S) | | | ✓ | <b>✓</b> | ✓ | ✓ | ✓ | ✓ | <b>~</b> | ✓ |

R : spécifique à la recherche,

S : spécifique aux Soins

(\*) AvAP : avant aph rèse / AvLD : avant lymphodépletion

Version n°2 du 08.10.2025 CONFIDENTIEL Page **27** sur **54** 





# 7.3 Visite de pré-inclusion/inclusion

# 7.3.1 Information Patient

Lors de la visite de pré-inclusion/inclusion, le médecin investigateur informera le participant et répondra à toutes ses questions concernant l'objectif, la nature des contraintes, les risques prévisibles et les bénéfices attendus de l'étude clinique. Il précisera également les droits du participant dans le cadre d'une recherche et vérifiera les critères d'éligibilité.

L'investigateur laissera au patient un délai de réflexion de minimum 30 minutes.

# 7.3.2 Recueil du consentement

Après vérification des critères d'éligibilité, le médecin investigateur sera responsable de l'obtention du consentement du patient.

Le patient et l'investigateur inscriront leurs noms et prénoms en clair, dateront et signeront le formulaire de consentement avant toute prémédication susceptible d'altérer la vigilance du patient. Celui-ci <u>doit</u> <u>être signé avant la réalisation de tout examen</u> clinique ou biologique ou para-clinique nécessité par la recherche.

L'exemplaire <u>original</u> sera conservé dans le dossier informatique du patient. Un exemplaire (un autre original ou une copie) sera remis au patient.

L'investigateur précisera dans le dossier médical du patient sa participation à la recherche, les modalités du recueil du consentement ainsi que celle de l'information.

# 7.3.3 Déroulement de la visite – V0 (AvAP)

La visite de pré-inclusion/inclusion est assurée par le médecin investigateur, et suit les procédures en vigueur pour les patients recevant un CAR-T.

#### Seront réalisés:

- Un examen clinique (selon les pratiques usuelles du suivi de leur pathologie et pour traitement par cellules CART-BCMA),
- Un prélèvement sanguin, si nécessaire pour le suivi habituel de leur pathologie, auquel sera couplé un prélèvement d'environ 25mL de sang supplémentaires pour l'étude, si tel n'est pas le cas il aura un prélèvement spécifique pour cette étude.

Pour la recherche, des données seront recueillies dans le dossier médical du patient :

- Age, sexe,
- Type immunoglobine monoclonale (IgA, IgD, IgG, kappa, lamba, non-secretory),
- Pourcentage d'infiltration plasmocytaire dans la MO,
- ISS et R-ISS stages,
- Risques cytogénétiques sur moelle osseuse,
- Rechutes du MM et lignes thérapeutiques précédentes,
- Délai entre diagnostic et la thérapie CAR-T,
- Type de CAR-T : IdeCel/cilta cell, traitement d'attente
- Obtention d'une rémission complète ou non (répondeur ou non au traitement par CART),
- Traitements reçus pendant le délai de production des CAR-BCMA (entre les visites V0 et V1),

Version n°2 du 08.10.2025 CONFIDENTIEL Page **28** sur **54** 





- Traitement par greffe autologue de cellules souches, avant le traitement par CAR-BCMA.

# 7.4 Visites de suivi

# Visite V1: avant lymphodéplétion, 6 à 8 semaines après la visite d'inclusion/aphérèse V0,

- Un examen clinique (selon les pratiques usuelles du suivi de leur pathologie),
- Un prélèvement sanguin, si nécessaire pour le suivi habituel de leur pathologie, auquel sera couplé un prélèvement d'environ 25mL supplémentaires pour l'étude, si tel n'est pas le cas il aura un prélèvement spécifique pour cette étude,
- Un prélèvement médullaire nécessaire pour le suivi habituel de leur pathologie, auquel sera couplé un prélèvement de 3 à 5 mL supplémentaires pour l'étude.

# Visite V2 : J10 soit 10 jours après infusion du produit CART

- Un examen clinique (selon les pratiques usuelles du suivi de leur pathologie),
- Un prélèvement sanguin, si nécessaire pour le suivi habituel de leur pathologie, auquel sera couplé un prélèvement d'environ 25mL supplémentaires pour l'étude, si tel n'est pas le cas il aura un prélèvement spécifique pour cette étude.

# Visite V3: M1 soit un mois après infusion du produit CART

- Un examen clinique (selon les pratiques usuelles du suivi de leur pathologie),
- Un prélèvement sanguin, si nécessaire pour le suivi habituel de leur pathologie, auquel sera couplé un prélèvement d'environ 25mL supplémentaires pour l'étude, si tel n'est pas le cas il aura un prélèvement spécifique pour cette étude.

# Visite V4 : M3 soit 3 mois après infusion du produit CART

- Un examen clinique (selon les pratiques usuelles du suivi de leur pathologie),
- Un prélèvement sanguin, si nécessaire pour le suivi habituel de leur pathologie, auquel sera couplé un prélèvement d'environ 25mL supplémentaires pour l'étude, si tel n'est pas le cas il aura un prélèvement spécifique pour cette étude,
- Un prélèvement médullaire nécessaire pour le suivi habituel de leur pathologie, auquel sera couplé un prélèvement de 3 à 5 mL supplémentaires pour l'étude.

# <u>Visite V5 : M6 soit 6 mois après infusion du produit CART</u>

- Un examen clinique (selon les pratiques usuelles du suivi de leur pathologie),
- Un prélèvement sanguin, si nécessaire pour le suivi habituel de leur pathologie, auquel sera couplé un prélèvement d'environ 25mL supplémentaires pour l'étude, si tel n'est pas le cas il aura un prélèvement spécifique pour cette étude.

# Visite V6: M12 soit 12 mois après infusion du produit CART

- Un examen clinique (selon les pratiques usuelles du suivi de leur pathologie),
- Un prélèvement sanguin, si nécessaire pour le suivi habituel de leur pathologie, auquel sera couplé un prélèvement d'environ 25mL supplémentaires pour l'étude, si tel n'est pas le cas il aura un prélèvement spécifique pour cette étude
- Un prélèvement médullaire nécessaire pour le suivi habituel de leur pathologie, auquel sera couplé un prélèvement de 3 à 5 mL supplémentaires pour l'étude

Les prélèvements recueillis lors des visites de suivis sont destinés aux immunophénotypages et à l'analyse de facteurs solubles.

Version n°2 du 08.10.2025 CONFIDENTIEL Page **29** sur **54** 





Pour la recherche, des données seront recueillies à chaque visite dans le dossier médical du patient :

- Statut répondeur / non-répondeur données cliniques associées
- Obtention d'une rémission complète ou non suivant les IMWG

# 7.5 Visite de Suivi FU

Visite de FU 1 : 6 mois post M12 et Visite FU2 :12 mois post M12

- Evolution de la réponse au traitement depuis le M12 suivant les IMWG

# 7.6 Règles d'arrêt

# 7.6.1 <u>de la participation d'une personne</u>

L'investigateur pourra interrompre définitivement la participation d'un patient à l'étude pour toute raison qui servirait au mieux les intérêts du patient comme par exemple :

- Retrait de consentement en cours d'étude : les patients peuvent retirer leur consentement et demander à sortir de l'étude à n'importe quel moment et ce, quelle qu'en soit la raison,
- Toute raison qui servirait au mieux les intérêts du sujet (par exemple en cas d'événements indésirables graves nécessitant une prise en charge incompatible avec le protocole).

La date et la raison de la sortie d'essai devront être notées dans le dossier médical du patient et le cahier d'observation.

Le patient qui choisit d'abandonner ou de retirer son consentement ne bénéficiera plus d'aucune procédure d'étude dans le cadre du protocole. Les soins standards seront effectués selon les meilleures pratiques cliniques compte tenu de son état de santé.

Le patient qui choisit de retirer son consentement n'aura plus de données supplémentaires collectées et sera considéré comme perdu de vue dans l'analyse de survie. Tout échantillon biologique lui appartenant sera détruit à sa demande.

Le patient qui ne termine pas la visite 6 (en dehors du décès) et qui choisit d'abandonner ou de retirer son consentement sera remplacé.

L'investigateur doit identifier la cause de l'abandon si possible et évaluer s'il est possible de collecter la variable sur laquelle porte le critère d'évaluation principal au moment de l'abandon. Les abandons de recherche doivent être notifiés rapidement au site coordinateur et au promoteur par télécopie. Toutes les données obtenues entre la date de signature du formulaire de consentement éclairé et la date d'abandon resteront évaluables aux fins de l'étude.

Les raisons et la date de l'abandon pour le patient qui choisit d'abandonner, doivent être documentées dans le dossier du patient ainsi que le refus de consentement au traitement des données supplémentaires collectées dans le cadre de l'étude.

#### 7.6.2 *De l'étude*

L'étude se terminera normalement comme prévu dans le protocole. Le promoteur se réserve le droit d'interrompre l'étude à tout moment, notamment si les objectifs d'inclusion ne sont pas remplis.

Version n°2 du 08.10.2025 CONFIDENTIEL Page 30 sur 54





La survenue de certains faits pourra entraîner une suspension temporaire ou une fin anticipée de l'étude clinique.

# 7.7 <u>Contraintes liées à l'étude clinique et indemnisation éventuelle des participants</u>

La personne peut participer à une autre recherche, à l'exception de celle(s) nécessitant une prise de sang et faisant alors dépasser le volume total maximal de sang prélevé dans les 4 semaines précédant ou suivant la présente étude, en accord avec l'arrêté du 12/04/2018 fixant la liste des recherches mentionnées au 2° de l'article L. 1121-1 du code de la santé publique.

Cette étude ne nécessitant aucun déplacement spécifique pour les patients, ils ne percevront pas d'indemnité de déplacement.

# 7.8 <u>Inscription du participant de l'étude clinique dans le fichier national des personnes qui se prêtent à des recherches</u>

Non applicable

Version n°2 du 08.10.2025 CONFIDENTIEL Page **31** sur **54** 





# 8 PROCEDURE ET STRATEGIES

# 8.1 Analyse cellulaire des prélèvements de sang total et de moelle osseuse

Les méthodes utilisées sont principalement celles de l'immunologie cellulaire chez l'humain comprenant des analyses phénotypiques adaptés à la nouvelle technologie de cytométrie en flux multiparamétrique spectrale (CFMS) comprenant la validation d'un nouveau panel de marquage (35 marqueurs analysés simultanément).

A cette fin, nous utiliserons le cytomètre spectral Aurora (Cytek) de la plateforme de cytométrie en flux de l'Université de Poitiers.

Après décongélation, immunomarquage extra et intracellulaire, puis acquisition, les données de cytométrie en flux seront analysées avec le logiciel FlowJo v10 (BD Biosciences).

L'analyse des populations de lymphocytes étant réalisée sur des cellules congelées, il est important de noter que nos travaux antérieurs ont validé l'absence de biais significatif dans l'analyse des phénotypes et des fonctions en lien avec la congélation des échantillons de cellules sanguines et de MO. Après décongélation des échantillons et immuno-marquage membranaire de surface et intracellulaire (cytoplasmique (perforine, granzymes) et nucléaire (facteurs de transcription)), les CMN seront analysées simultanément pour 36 paramètres de fluorescence à partir d'un unique panel d'immuno-marquage.

Notre stratégie d'analyse consistera à employer le pipeline suivant (Liechti et al. 2021; Rybakowska et al. 2020):

- 1) création de panels multiparamétriques optimisés et utilisation d'un protocole standardisé de marquage cellulaire
- 2) acquisition des données sur le cytomètre spectral
- 3) Déconvolution spectrale (unmixing) et éventuelles compensations corrigeant les erreurs de l'algorithme de déconvolution
- 4) normalisation des données et si nécessaire correction des batch-effects.

Enfin, les données seront analysées de façon supervisée et non-supervisées tel que décrit cidessous.

# 8.2 <u>Analyses supervisées</u>

Les cellules seront analysées par CFMS dans une fenêtre de CMN excluant les débris et les cellules mortes (LiveDead négative).

Dans un premier temps, les celllules CAR-T positives seront identifiées par marquage au BCMA-biotinylé avec détection par un anticorps secondaire anti-biotin couplé à la PE.

Dans les deux sous-populations ainsi identifiées (CAR-T(+) et CAR-T(-)), les populations immunitaires d'intérêt seront identifiées selon les critères phénotypiques suivants :

- 1) iNKT : CD3(+) et anticorps clone 6B11(+) spécifique de la région jonctionnelle  $V\alpha 24$ -Ja18 du TCR des iNKT.
- 2) MAIT : CD161(+) TCR  $V\alpha7.2(+)$  parmi les cellules CD3(+),
- 3) LT-V $\delta$ 1 et LT $\delta$ 2 : CD3(+) TCR-V $\delta$ 1(+) ou TCR-V $\delta$ 2(+),
- 4) Les LTI CD8 : définis par l'expression d'un des récepteurs suivants KIR3DL1/DL2, PanKir2D, NKG2A parmi les LT CD8(+) et après exclusion des iNKT, MAIT et LT- $\gamma\delta$ ,

Version n°2 du 08.10.2025 CONFIDENTIEL Page **32** sur **54** 





- **5**) Les LT conventionnels (conv) T CD8(+) et T CD4(+) dans une fenêtre d'exclusion des LTI CD8 et des Treg et des Treg respectivement,
- 6) Les LT CD4(+) Treg : CD4(+) FoxP3(+) CD25(+).

Nous déterminerons en premier lieu la fréquence et le nombre absolu des iNKT, MAIT, LTI CD8, LT-γδ, Treg, LT CD4conv et LT CD8conv au sein des cellules CAR-T(+) et CAR-T(-).

Pour chacune des sous-populations identifiées, nous analyserons les marqueurs phénotypiques suivants : CD45RA, CCR7, CD28, CD62L, CXCR3, CD69, CD137, TIGIT, PD-1, CD122, Eomes, Helios, T-bet, PLZF, TCF-1, CD95, CD95L, perforine, granzyme et Ki67.

# 8.3 Analyses non supervisées

Après nettoyage des données décrit ci-dessus, le pipeline suivant sera utilisé :

- 1) la réduction de dimensions (algorithmes tels que UMAP, Opt-SNE) pour obtenir une carte en 2D interprétable par l'oeil humain et reflétant tous les paramètres étudiés, puis
- 2) l'utilisation d'algorithmes de classifications (clustering tels que FlowSOM, PhenoGraph) pour identifier les différentes populations cellulaires aux caractéristiques différentes ;
- 3) des statistiques descriptives, d'analyses de différences et de prédiction seront ensuite appliquées pour identifier les variations de population ou d'expression de marqueurs d'intérêt, enfin
- 4) les résultats obtenus seront vérifiés par une stratégie d'analyse manuelle dirigée.

# 8.4 <u>Dosages cytokiniques des sérums</u>

Les tubes secs (rouges) collectés à chaque prélèvement de sang total seront centrifugés 15 min à 2000 g et les surnageants seront aliquotés et conservés à -80°C.

Le dosage des cytokines pro-inflammatoires sera réalisé au laboratoire d'immunologie clinique (Pr. Jean-Marc GOMBERT) du CHU de Poitiers, par la méthode/automate Ella (Protein Simple) après décongélation et dilution du sérum.

Les cytokines IL-1 $\beta$ , IFN- $\gamma$ , IL-6, IL-10, IL-15 et TNF- $\alpha$  seront dosées avec des cartouches en simplex ou en multiplex.

Le dosage de sCD95L sera réalisé par méthode ELISA (Abcam Human FAS Ligand (CD95L) ELISA kit, #AB45892) dans l'équipe du Dr Patrick LEGEMBRE (DR INSERM, Limoges) après décongélation, selon les recommandations du fournisseur.

Les résultats des dosages de chaque cytokine à chaque temps du suivi longitudinal, seront corrélés au pourcentage des LT CART-BCMA déterminé par cytométrie en flux spectrale.

Version n°2 du 08.10.2025 CONFIDENTIEL Page **33** sur **54** 





# 9 COLLECTION D'ECHANTILLONS BIOLOGIQUES

# 9.1 <u>Description des collections</u>

# 9.1.1 Sang et sérum:

20 mL de sang périphérique en tubes EDTA et un tube de 5 mL de sang périphérique en tube sec CAT prélevés par ponction veineuse aux visites :

- Inclusion, avant aphérèse (V0),
- Avant la lymphodéplétion (V1),
- À J10 après l'injection du produit CAR-T cells (V2),
- À M1 après l'injection du produit CAR-T cells (V3),
- À M3 après l'injection du produit CAR-T cells (V4),
- À M6 après l'injection du produit CAR-T cells (V5),
- À M12 après l'injection du produit CAR-T cells (V6),

A l'issue de la recherche, un aliquot des échantillons de sérums de chaque patient seront envoyés par transporteur en carboglace au laboratoire CRIBL à l'Université de Limoges (sous la responsabilité du Dr. Patrick LEGEMBRE et du Dr. Murielle ROUSSEL) pour effectuer les dosages du CD95L solubles et autres cytokines d'intérêt.

# 9.1.2 Moelle osseuse

3 à 5 mL de moelle osseuse en tubes EDTA. Le prélèvement de moelle osseuse s'effectue sous anesthésie locale, au niveau du sternum ou de l'os de la hanche avec un trocart, sur lequel est adaptée une seringue pour aspirer la moelle osseuse, aux visites :

- Avant la lymphodéplétion (V1),
- À M3 après l'injection du produit CAR-T cells (V4),
- À M12 après l'injection du produit CAR-T cells (V6),

Les tubes seront identifiés avec les étiquettes fournies : nom de l'étude (CART-I5M/PBS-IRATI), numéro du patient suivi la visite correspondante (inclusion, V2...) et la fiche de prélèvement sera complétée.

Les prélèvements accompagnés de la fiche de prélèvement seront envoyés au Centre de Ressources Biologiques du CHU de Poitiers afin de réaliser la mise en conformité, pseudonymisation et traçabilité.

Les 20 mL de sang périphérique et les 5 mL de moelle osseuse en tubes EDTA seront immédiatement transférés au laboratoire d'immunologie de l'unité INSERM U1313.

Les cellules mononucléées (CMN) et le plasma seront dès lors séparées du sang total par centrifugation en gradient de densité sur une solution de Ficoll.

Les CMN seront congelées et stockées dans l'azote liquide au sein du laboratoire, les plasmas seront aliquotés (3\*500µL) et congelés à -80°C.

Les sérums seront séparés par centrifugation, aliquotés (3\*500µL) et congelés à -80°C.





Après décongélation et immunomarquages extra et intracellulaire, les CMN seront analysées à l'aide d'un cytomètre multiparamétrique spectral (Aurora spectral analyzer, Cytek) et les données avec les logiciels FlowJo v10 (Treestar.Inc).

Les plasmas seront analysés par des techniques de dosages de protéines par ELISA ou autre technique à haut débit.

# 9.2 Transports

Les échantillons seront acheminés du CRB au laboratoire INSERM U1313 de l'Université de Poitiers, à température ambiante via la navette prévue à cet effet, dans un délai n'excédant pas 24 heures de transport.

Dans ces conditions, la qualité du prélèvement n'est pas compromise comme cela a été éprouvé à travers nos projets antérieurs.

# 9.3 Conservation

Les échantillons seront conservés de manière transitoire (moins de 24h) au sein du CRB du CHU de Poitiers, entrée 5 cour Est Jean-Bernard, 2 rue de la Milétrie, 86021 Poitiers cedex.

Les échantillons seront conservés et analysés au sein du laboratoire INSERM U1313, B36 Université de Poitiers, 1 rue Georges Bonnet, 86000 Poitiers.

Les CMN de sang périphérique et de moelle osseuse seront stockées dans l'azote liquide (-170°C), les plasmas seront aliquotés (3x500μL) et congelés à -80°C au sein du laboratoire INSERM U1313.

### 9.4 Devenir de la collection

Pendant la recherche, la collection d'échantillons biologiques sera conservée par l'équipe INSERM U1313 sous la responsabilité du Dr BOBIN Arthur jusqu'à la fin de la recherche.

Le CRIBL de l'Université de Limoges détruira le sérum potentiellement restant après analyse. Aucune collection biologique au CRIBL de l'Université de Limoges n'est prévu.

A l'issue de la recherche, les échantillons restants au laboratoire INSERM U1313 de Poitiers seront utilisés pour des analyses ultérieures concernant le MM non prévues dans le protocole pouvant se révéler intéressantes en fonction de l'évolution des connaissances scientifiques, sous réserve que le participant n'y soit pas opposé, après en avoir été informé, comme indiqué dans la note d'information/consentement.

La collection sera déclarée au ministre chargé de la recherche et au directeur de l'agence régionale de santé territorialement compétent (article L. 1243-3 du CSP).

Version n°2 du 08.10.2025 CONFIDENTIEL Page 35 sur 54



CART-I5M

| Type de<br>prélèvement | Lieu<br>conservation | Responsable de la collection | Finalité de<br>la collection | Durée de la conservation | Devenir |
|---|---|---|---|---|---|
| Sanguins | INSERM<br>U1313 | Dr BOBIN Arthur | Recherche | Epuisement de la collection | Epuisement |
| Moelle<br>osseuse | INSERM<br>U1313 | Dr BOBIN Arthur | Recherche | Epuisement de la collection | Epuisement |




# 10 GESTION DES EVENEMENTS INDESIRABLES / EFFETS INDESIRABLES / INCIDENTS

Les évènements indésirables / effets indésirables / incidents seront à déclarer aux différents circuits de vigilances sanitaires applicables à chaque produit ou pratique concernée (vigilance du soin, pharmacovigilance, hémovigilance, cosmétovigilance...) en conformité avec la règlementation en vigueur.

Les déclarants doivent spécifier que la patiente est incluse dans un essai clinique et identifier précisément l'essai clinique concerné.

Si l'investigateur a connaissance d'une atteinte à la sécurité des patientes dans le cadre de la recherche, il doit en informer sans délai le promoteur.





## 11 ASPECTS STATISTIQUES

## 11.1 Calcul de la taille d'étude

Cette demande de collection biologique s'intègre dans le cadre de la recherche exploratoire à visée fondamentale, avec pour objectif principal de tester la corrélation de l'expression du facteur de transcription TCF-1 avec la persistance des cellules CART-BCMA.

En se basant sur de précédentes expérimentations de détection du facteur de transcription TCF-1, et le décroit rapide des cellules CART au cours du temps (détectable chez 1 patient sur 2 sur quelques microlitres de sang périphérique 3 mois après la réinjection), l'inclusion de 40 patients analysables au total, est nécessaire afin de garantir la qualité statistique des données obtenues.

Le CHU traite environ 1 à 2 patients atteints de MM par mois par thérapie CART-BCMA, l'objectif d'un recrutement de 40 patients analysables pour **60** incluables.

Ces effectifs seront suffisants pour pouvoir réaliser des t-test et des études d'associations clinicobiologiques.

Les analyses statistiques seront effectuées par le logiciel GrapPad Prism v10

## 11.2 Méthodes statistiques employées

Méthodes descriptives usuelles (moyenne, écart type, fréquence).

Les comparaisons de moyennes seront réalisées par un t test de de Student et les comparaisons de fréquence par la méthode du chi² d'indépendance. Les données non normalement distribuées seront analysées par un test de Mann-Whitney U pour les variables quantitatives.

Les études de corrélations seront évaluées par les coefficients de corrélation de Spearman pour les variables quantitatives.

Toutes les analyses seront réalisées avec un risque alpha bilatéral de 0,05.

Il n'y aura pas d'analyses intermédiaires.

Les analyses seront menées sous GraphPad PrismV10 (GraphPad Software, San Diego California, USA) et SASv9.4 (NYC, CAL)





# 12 GESTION ET TRAITEMENT DES DONNEES ET DOCUMENTS SOURCE

## 12.1 Données et documents source

Les données source correspondent à l'ensemble des informations figurant dans des documents originaux, ou dans des copies authentifiées de ces documents, relatif aux examens cliniques, aux observations ou à d'autres activités menées dans le cadre d'une recherche et nécessaires à la reconstitution et à l'évaluation de l'étude clinique.

Les documents dans lesquels les données sources sont enregistrées sont appelés les documents sources.

Les données nécessaires à la réalisation de la recherche sont saisies à partir du dossier médical du patient qui constitue le dossier source.

Les données sources (dossier médical, résultats d'examens, etc) sont conservées par l'investigateur qui s'engage à autoriser un accès direct aux données sources de l'étude clinique lors des visites de contrôle, d'audit ou d'inspection.

Les données suivantes seront relevées :

- âge, sexe,
- myélome : type d'immunoglobuline monoclonale impliquée, pourcentage d'infiltration plasmocytaire dans la MO, stade selon les classifications DS et ISS, risque cytogénétique),
- lignes thérapeutiques : traitement avant entrée dans le protocole, traitement reçu entre l'aphérèse et la lymphodéplétion)
- CAR-T :type de CART, répondeur/non répondeur
- survie.

Uniquement les données utiles à cette recherche seront collectées. Les données collectées seront analysées et seront décrites dans la publication de ce projet de recherche. Aucune autre donnée ne sera relevée.

## 12.2 Consignes pour le recueil des données

Toutes les informations requises par le protocole doivent être consignées sur les cahiers d'observation et une explication doit être apportée pour chaque donnée manquante. Les données doivent être recueillies au fur et à mesure qu'elles sont obtenues, et transcrites dans ces cahiers de façon nette et lisible.

Les données seront recueillies sur un cahier d'observation électronique (e-CRF)

Les données enregistrées dans l'e-CRF et provenant des documents sources doivent être cohérentes entre elles ; dans le cas contraire, les différences doivent être justifiées et documentées.

L'investigateur est responsable de l'exactitude, de la qualité et de la pertinence de toutes les données saisies.

Version n°2 du 08.10.2025 CONFIDENTIEL Page **39** sur **54** 





## 12.3 Gestion et circuit des données

L'e-CRF est développé, codé et mis en production par la plateforme Méthodologie-Biostatistiques et Data-Management du CHU de Poitiers, localisée à la Direction de la Recherche du CHU de Poitiers. La conception est réalisée par les data-managers.

L'équipe de Data-Management du CHU de Poitiers octroie les droits d'accès des personnes qui ont été identifiées pour saisir et valider dans l'e-CRF par site.

Le cahier d'observation électronique disponible dans le centre via internet et un lien vers le module de recueil de données.

De plus, lors de leurs saisies, ces données sont immédiatement vérifiées grâce à des contrôles de cohérence (A ce titre, l'investigateur doit valider toute modification de valeur dans le CRF.). Ces modifications font l'objet d'un audit trail. Une justification peut éventuellement être intégrée en commentaire.

Une copie e-CRF sous format PDF de chaque participant complété par centre et authentifié par le promoteur sera envoyé au centre participant via un CD/CD/ROM et devra être archivée par l'investigateur de chaque centre participant.

## 12.4 <u>Confidentialité des données</u>

Conformément aux dispositions législatives en vigueur, les personnes ayant un accès direct aux données source prendront toutes les précautions nécessaires en vue d'assurer la confidentialité des informations relatives aux médicaments expérimentaux, aux recherches, aux personnes qui s'y prêtent et notamment en ce qui concerne leur identité ainsi qu'aux résultats obtenus.

Ces personnes, au même titre que les investigateurs eux-mêmes, sont soumises au secret professionnel.

Pendant la recherche ou à son issue, les données recueillies sur les personnes qui s'y prêtent et transmises au promoteur par les investigateurs (ou tous autres intervenants spécialisés) seront rendues anonymes. Elles ne doivent en aucun cas faire apparaître en clair les noms des personnes concernées ni leur adresse.

Seules les initiales du nom et du prénom du patient seront enregistrées, accompagnées d'un numéro codé propre à l'étude indiquant l'ordre d'inclusion des sujets.

Le promoteur s'assurera que chaque personne qui se prête à la recherche a donné son accord par écrit pour l'accès aux données individuelles la concernant et strictement nécessaires au contrôle de qualité de la recherche.

Une liste de correspondance sera conservée par l'investigateur principal du centre participant dans le classeur de l'étude clinique. Cette liste de correspondance fait partie des documents de l'étude clinique et sera conservée pour une durée de 15 ans après la fin de la recherche.

Aucune information permettant l'identification des participants ne sera communiquée à des tiers, représentants du promoteur et aux autorités compétentes, réglementairement habilitées à détenir cette information et qui sont tous tenus au secret professionnel.

Version n°2 du 08.10.2025 CONFIDENTIEL Page **40** sur **54** 





## 12.5 Conservation des documents et des données relatifs à l'étude

Les documents suivants relatifs à cette recherche sont archivés par l'investigateur conformément aux Bonnes Pratiques Cliniques, à l'arrêté du 11 août 2008 fixe la durée de conservation des documents relatifs aux recherches en santé:

- pour une durée de 15 ans suivant la fin de la recherche (recherches ne portant pas sur un produit mentionné à l'article L.5311-1 du code de la santé publique),
  - Le protocole et les modifications éventuelles au protocole
  - Les cahiers d'observation (copies)
  - Les dossiers source des participants ayant signé un consentement
  - Tous les autres documents et courriers relatifs à la recherche
  - L'exemplaire original des consentements signés des participants

Tous ces documents sont sous la responsabilité de l'investigateur pendant la durée réglementaire d'archivage.

Aucun déplacement ou destruction ne pourra être effectué sans l'accord du promoteur. Au terme de la durée réglementaire d'archivage, le promoteur sera consulté pour destruction. Toutes les données, tous les documents et rapports pourront faire l'objet d'audit ou d'inspection.

Les données recueillies pour l'étude seront accessibles aux personnes habilitées par le CHU de Poitiers, pendant deux ans après la dernière publication des résultats de la recherche. Elles feront l'objet d'un archivage pendant 15 ans après la fin de l'étude conformément à la réglementation en vigueur.

## 12.6 Cession des données

La gestion des données est assurée par le CHU de Poitiers.

Les conditions de cession de tout ou partie de la base de données de l'étude clinique sont décidées par le promoteur de l'étude clinique et font l'objet d'un contrat écrit au préalable.





## 13 CONTROLE ET ASSURANCE QUALITE

## 13.1 Accès aux données

L'acceptation de la participation au protocole implique que les investigateurs mettront à disposition les documents et données individuelles strictement nécessaires au suivi, au contrôle de qualité et à l'audit de l'étude clinique, à la disposition des personnes ayant un accès à ces documents conformément aux dispositions législatives et réglementaires en vigueur.

## 13.2 Contrôle Qualité

Un attaché de recherche clinique mandaté par le promoteur visite le site investigateur conformément au plan de monitorage basé sur le risque (participant, logistique, impact, ressources), au minimum les éléments suivants seront revus le Consentement des patients, le respect du protocole de l'étude clinique. Toute visite fera l'objet d'un rapport de monitorage par compte-rendu écrit.

## 13.3 Audit et inspections

Un audit peut être réalisé à tout moment par des personnes mandatées par le promoteur et indépendantes des personnes menant l'étude clinique. Il a pour objectif de vérifier la sécurité des participants et le respect de leurs droits, le respect de la réglementation applicable et la fiabilité des données.

Une inspection peut également être diligentée par une autorité compétente (ANSM pour la France ou EMA dans le cadre d'un essai européen par exemple).

L'audit, aussi bien que l'inspection, pourront s'appliquer à tous les stades de l'étude clinique, du développement du protocole à la publication des résultats et au classement des données utilisées ou produites dans le cadre de l'étude clinique.

Les investigateurs acceptent de se conformer aux exigences du promoteur en ce qui concerne un audit et à l'autorité compétente pour une inspection de l'étude clinique.





## 14 CONSIDERATIONS ETHIQUES ET REGLEMENTAIRES

Le promoteur et l'(es) investigateur(s) s'engagent à ce que cette recherche soit réalisée en conformité avec la loi n°2012-300 du 5 mars 2012 relative aux recherches impliquant la personne humaine/le Règlement Européen n°536/2014 du 16 avril 2014 relatif aux essais cliniques de médicaments, ainsi qu'en accord avec les Bonnes Pratiques Cliniques et les I.C.H. en vigueur et la déclaration d'Helsinki (qui peut être retrouvée dans sa version intégrale sur le site <a href="http://www.wma.net">http://www.wma.net</a>).

L'étude clinique est conduite conformément au présent protocole. Hormis dans les situations d'urgence nécessitant la mise en place d'actes thérapeutiques précis, l'(es) investigateur(s) s'engage(nt) à respecter le protocole en tous points en particulier en ce qui concerne le recueil du consentement.

#### CPP/ANSM:

L'étude clinique a été étudié et a reçu l'avis favorable du Comité de Protection des Personnes Ile de France IV (CPP IDF IV)

Le CHU de Poitiers transmettra l'avis favorable du CPP ainsi que le résumé du protocole à l'Agence Nationale de Sécurité du Médicaments et des produits de santé (ANSM).

#### Assurance:

Le CHU de Poitiers, promoteur de cette recherche, a souscrit un contrat d'assurance en responsabilité civile auprès de HDI Global SE (Tour Trinity, 1 bis place de la Défense, CS 20298, 92035 La Défense Cedex- Tel 01.44.06.56.00), contrat d'assurance n°7666522730013, conformément aux dispositions de l'article L1121-10 du code de la santé publique.

#### CNIL/RGPD:

Les données enregistrées à l'occasion de cette recherche font l'objet d'un traitement informatisé par le promoteur dans le respect de la loi n°78-17 du 6 janvier 1978 relative à l'informatique, aux fichiers et aux libertés modifiée par la loi 2004-801 du 6 août 2004 et la loi n°2018-493 du 20 juin 2018 relative à la protection des données personnelles;.

L'étude respectera le Règlement Général sur la Protection des Données (RGPD) n°2016-679 du 27 avril 2016.

Cette recherche entre dans le cadre de la « Méthodologie de référence » (MR-001) homologuée par délibération n°2018-153 du 3 mai 2018, entrée en vigueur le 13 juillet 2018. Le CHU de Poitiers a signé un engagement de conformité à cette « Méthodologie de référence ».

Cette étude clinique est enregistrée sur le site http://clinicaltrials.gov/

#### Modifications au protocole :

Toute modification substantielle, c'est à dire toute modification de nature à avoir un impact significatif sur la protection des personnes, sur les conditions de validité et sur les résultats de l'étude clinique, sur la qualité et la sécurité des produits expérimentés, sur l'interprétation des documents scientifiques qui viennent appuyer le déroulement de l'étude clinique ou sur les modalités de conduite de celle-ci, fait l'objet d'un amendement écrit qui est soumis au promoteur ; celui-ci doit obtenir, préalablement à sa mise en œuvre, un avis favorable du CPP.

Les modifications non substantielles, c'est à dire celles n'ayant pas d'impact significatif sur quelque aspect de l'étude clinique que ce soit, sont communiquées au CPP à titre d'information.

Version n°2 du 08.10.2025 CONFIDENTIEL Page 43 sur 54





Toutes les modifications sont validées par le promoteur, et par tous les intervenants de l'étude clinique concernés par la modification, avant soumission au CPP. Cette validation peut nécessiter la réunion de tout comité constitué pour l'étude clinique.

Toutes les modifications au protocole doivent être portées à la connaissance de tous les investigateurs qui participent à l'étude clinique. Les investigateurs s'engagent à en respecter le contenu.

Toute modification qui modifie la prise en charge des participants ou les bénéfices, risques et contraintes de l'étude clinique fait l'objet d'une nouvelle note d'information et d'un nouveau formulaire de consentement dont le recueil suit la même procédure que celle précitée.





## 15 REGLES RELATIVES A LA PUBLICATION

## 15.1 <u>Communications scientifiques</u>

L'analyse des données fournies par le centre investigateur sera réalisée par l'équipe de l'unité U1313 de l'Université de Poitiers en collaboration avec l'investigateur coordonnateur.

Cette analyse donnera lieu à un rapport écrit qui sera soumis au promoteur, qui le transmettra au Comité de Protection des Personnes.

Toute communication écrite ou orale des résultats de l'étude clinique doit recevoir l'accord préalable de l'investigateur coordonnateur et, le cas échéant, de tout comité constitué pour l'étude clinique. Un export partiel des données pseudonymisées descriptives pourra être réalisé au cours de la recherche dans le cadre de communication ou poster.

L'investigateur coordonnateur/principal s'engage à mettre à disposition du public les résultats de l'étude clinique aussi bien négatifs et non concluants que positifs.

La publication des résultats principaux mentionne le nom du CHU de Poitiers, de tous les investigateurs ayant inclus ou suivi des participants dans l'étude clinique, et les sources de financement.

Il sera tenu compte des règles internationales d'écriture et de publication (*The Uniform Requirements for Manuscripts* de l'ICMJE, avril 2010).

## 15.2 Communication des résultats aux participants

Conformément à la loi n°2002-303 du 4 mars 2002, les participants sont informés, à leur demande, des résultats globaux de l'étude clinique.





# 16 RÉFÉRENCES BIBLIOGRAPHIQUES

- Abken, Hinrich. 2016. "Costimulation Engages the Gear in Driving CARs." *Immunity* 44 (2): 214–16. https://doi.org/10.1016/j.immuni.2016.02.001.
- Alizadeh, Darya, Robyn A. Wong, Sharareh Gholamin, et al. 2021. "IFNγ Is Critical for CAR T Cell-Mediated Myeloid Activation and Induction of Endogenous Immunity." *Cancer Discovery* 11 (9): 2248–65. https://doi.org/10.1158/2159-8290.CD-20-1661.
- Brown, Christine E., and Crystal L. Mackall. 2019. "CAR T Cell Therapy: Inroads to Response and Resistance." *Nature Reviews. Immunology* 19 (2): 73–74. https://doi.org/10.1038/s41577-018-0119-y.
- Cazaux, Marine, Capucine L. Grandjean, Fabrice Lemaître, et al. 2019. "Single-Cell Imaging of CAR T Cell Activity in Vivo Reveals Extensive Functional and Anatomical Heterogeneity." *The Journal of Experimental Medicine* 216 (5): 1038–49. https://doi.org/10.1084/jem.20182375.
- Chang, Hyun-Dong, Koji Tokoyoda, and Andreas Radbruch. 2018. "Immunological Memories of the Bone Marrow." *Immunological Reviews* 283 (1): 86–98. https://doi.org/10.1111/imr.12656.
- Chen, Gregory M., Changya Chen, Rajat K. Das, et al. 2021. "Integrative Bulk and Single-Cell Profiling of Premanufacture T-Cell Populations Reveals Factors Mediating Long-Term Persistence of CAR T-Cell Therapy." *Cancer Discovery* 11 (9): 2186–99. https://doi.org/10.1158/2159-8290.CD-20-1677.
- Dimopoulos, M. A., P. Moreau, E. Terpos, et al. 2021. "Multiple Myeloma: EHA-ESMO Clinical Practice Guidelines for Diagnosis, Treatment and Follow-Up†." *Annals of Oncology* 32 (3): 309–22. https://doi.org/10.1016/j.annonc.2020.11.014.
- Dunn, Gavin P., Lloyd J. Old, and Robert D. Schreiber. 2004. "The Three Es of Cancer Immunoediting." *Annual Review of Immunology* 22: 329–60. https://doi.org/10.1146/annurev.immunol.22.012703.104803.
- Favreau, Mérédis, Koen Venken, Sylvia Faict, et al. 2017. "Both Mucosal-Associated Invariant and Natural Killer T-Cell Deficiency in Multiple Myeloma Can Be Countered by PD-1 Inhibition." *Haematologica* 102 (7): e266–70. https://doi.org/10.3324/haematol.2017.163758.
- Gattinoni, Luca, Enrico Lugli, Yun Ji, et al. 2011. "A Human Memory T Cell Subset with Stem Cell-like Properties." *Nature Medicine* 17 (10): 1290–97. https://doi.org/10.1038/nm.2446.
- Good, Charly R., M. Angela Aznar, Shunichiro Kuramitsu, et al. 2021. "An NK-like CAR T Cell Transition in CAR T Cell Dysfunction." *Cell* 184 (25): 6081-6100.e26. https://doi.org/10.1016/j.cell.2021.11.016.
- Kawalekar, Omkar U., Roddy S. O'Connor, Joseph A. Fraietta, et al. 2016. "Distinct Signaling of Coreceptors Regulates Specific Metabolism Pathways and Impacts Memory Development in CAR T Cells." *Immunity* 44 (2): 380–90. https://doi.org/10.1016/j.immuni.2016.01.021.
- Klebanoff, Christopher A., Christopher D. Scott, Anthony J. Leonardi, et al. 2016. "Memory T Cell-Driven Differentiation of Naive Cells Impairs Adoptive Immunotherapy." *The Journal of Clinical Investigation* 126 (1): 318–34. https://doi.org/10.1172/JCI81217.
- Kumar, Vivek, Neha Chaudhary, Mohit Garg, Charalampos S. Floudas, Parita Soni, and Abhinav B. Chandra. 2017. "Current Diagnosis and Management of Immune Related Adverse Events (irAEs) Induced by Immune Checkpoint Inhibitor Therapy." *Frontiers in Pharmacology* 8: 49. https://doi.org/10.3389/fphar.2017.00049.
- Liechti, Thomas, Lukas M. Weber, Thomas M. Ashhurst, et al. 2021. "An Updated Guide for the Perplexed: Cytometry in the High-Dimensional Era." *Nature Immunology* 22 (10): 1190–97. https://doi.org/10.1038/s41590-021-01006-z.





Page 47 sur 54

- Majzner, Robbie G., and Crystal L. Mackall. 2019. "Clinical Lessons Learned from the First Leg of the CAR T Cell Journey." *Nature Medicine* 25 (9): 1341–55. https://doi.org/10.1038/s41591-019-0564-6.
- Manier, Salomon, Tiziano Ingegnere, Guillaume Escure, et al. 2022. "Current State and Next-Generation CAR-T Cells in Multiple Myeloma." *Blood Reviews*, January 21, 100929. https://doi.org/10.1016/j.blre.2022.100929.
- Melenhorst, J. Joseph, Gregory M. Chen, Meng Wang, et al. 2022. "Decade-Long Leukaemia Remissions with Persistence of CD4+ CAR T Cells." *Nature* 602 (7897): 503–9. https://doi.org/10.1038/s41586-021-04390-6.
- Moreau, P., J. San Miguel, P. Sonneveld, et al. 2017. "Multiple Myeloma: ESMO Clinical Practice Guidelines for Diagnosis, Treatment and Follow-Up." *Annals of Oncology: Official Journal of the European Society for Medical Oncology* 28 (suppl\_4): iv52–61. https://doi.org/10.1093/annonc/mdx096.
- Munshi, Nikhil C., Jr Anderson Larry D., Nina Shah, et al. 2020. "Idecabtagene Vicleucel (Ide-Cel; Bb2121), a BCMA-Targeted CAR T-Cell Therapy, in Patients with Relapsed and Refractory Multiple Myeloma (RRMM): Initial KarMMa Results." *Journal of Clinical Oncology* 38 (15\_suppl): 8503–8503. https://doi.org/10.1200/JCO.2020.38.15\_suppl.8503.
- Rajkumar, S. Vincent. 2016. "Updated Diagnostic Criteria and Staging System for Multiple Myeloma." American Society of Clinical Oncology Educational Book. American Society of Clinical Oncology. Annual Meeting 35: e418-423. https://doi.org/10.1200/EDBK\_159009.
- Rybakowska, Paulina, Marta E. Alarcón-Riquelme, and Concepción Marañón. 2020. "Key Steps and Methods in the Experimental Design and Data Analysis of Highly Multi-Parametric Flow and Mass Cytometry." *Computational and Structural Biotechnology Journal* 18: 874–86. https://doi.org/10.1016/j.csbj.2020.03.024.
- Siegel, Rebecca L., Kimberly D. Miller, and Ahmedin Jemal. 2019. "Cancer Statistics, 2019." *CA: A Cancer Journal for Clinicians* 69 (1): 7–34. https://doi.org/10.3322/caac.21551.
- Yi, Fei, Tal Cohen, Natalie Zimmerman, et al. 2024. "CAR-Engineered Lymphocyte Persistence Is Governed by a FAS Ligand/FAS Auto-Regulatory Circuit." Preprint, bioRxiv, March 1. https://doi.org/10.1101/2024.02.26.582108.





### **ANNEXES**

Déclaration d'Helsinki de L'AMM - Principes éthiques applicables à la recherche médicale impliquant des êtres humains. Version Octobre 2024

#### **PRÉAMBULE**

1. L'Association médicale mondiale (AMM) a élaboré la Déclaration d'Helsinki comme un énoncé de principes éthiques applicables à la recherche médicale impliquant des participants humains, y compris la recherche utilisant du matériel humain ou des données personnelles identifiables.

La Déclaration est conçue comme un tout indissociable. Chaque paragraphe doit être appliqué en tenant compte de tous les autres paragraphes pertinents.

2. Bien que la Déclaration soit adoptée par les médecins, l'AMM considère que ces principes doivent être respectés par toutes les personnes, équipes et organisations impliquées dans la recherche médicale, car ils sont essentiels au respect et à la protection de tous les participants à la recherche, y compris les patients et les volontaires en bonne santé.

#### PRINCIPES GÉNÉRAUX

- 3. La Déclaration de Genève de l'AMM engage le médecin en ces termes : « La santé et le bien-être de mon patient [seront] ma priorité », et le Code international d'éthique médicale de l'AMM déclare « Le médecin doit s'engager à faire de la santé et du bien-être du patient sa priorité et à prodiguer ses soins dans l'intérêt supérieur de celui-ci ».
- 4. Le devoir du médecin est de promouvoir et de sauvegarder la santé, le bien-être et les droits des patients, y compris ceux des personnes impliquées dans la recherche médicale. Le médecin consacre son savoir et sa conscience à l'accomplissement de ce devoir.
- 5. Le progrès médical repose sur la recherche qui, en fin de compte, doit inclure des participants.

Même les interventions éprouvées devraient être évaluées en permanence par de la recherche portant sur leur sécurité, leur efficacité, leur pertinence, leur accessibilité et leur qualité.

- 6. La recherche médicale impliquant des participants humains est soumise à des normes éthiques qui promeuvent et garantissent le respect de tous les participants et protègent leur santé et leurs droits.
- La recherche médicale ayant lieu dans le contexte de diverses inégalités structurelles, les chercheurs devraient examiner attentivement la manière dont les bénéfices, les risques et les inconvénients sont répartis.
- Un engagement significatif avec les participants potentiels et inclus, et leurs communautés devrait se produire avant, pendant et après la recherche médicale. Les chercheurs doivent permettre aux participants potentiels et inclus, et à leurs communautés de partager leurs priorités et leurs valeurs, de participer à la conception et à la mise en œuvre de la recherche, ainsi qu'à d'autres activités pertinentes, et de s'engager dans la compréhension et la diffusion des résultats.
- 7. L'objectif premier de la recherche médicale impliquant des participants humains est de générer des connaissances pour comprendre les causes, le développement et les effets des maladies, d'améliorer les





interventions préventives, diagnostiques et thérapeutiques, et, en fin de compte, de faire progresser la santé individuelle et publique.

Ces objectifs ne peuvent jamais prévaloir sur les droits et intérêts des participants à la recherche.

- 8. Si de nouvelles connaissances et interventions peuvent s'avérer impérativement nécessaires en situation d'urgence de santé publique, il reste essentiel de respecter les principes éthiques énoncés dans la présente Déclaration lors de telles situations d'urgence.
- 9. Il est du devoir des médecins engagés dans la recherche médicale de protéger la vie, la santé, la dignité, l'intégrité, l'autonomie, la vie privée et la confidentialité des informations personnelles des participants impliqués dans la recherche. La responsabilité de protéger les participants à la recherche doit toujours incomber aux médecins ou aux autres chercheurs et jamais aux participants à la recherche, même s'ils ont donné leur consentement.
- 10. Les médecins et les autres chercheurs doivent tenir compte des normes et standards éthiques, légaux et réglementaires applicables à la recherche impliquant des participants humains dans le ou les pays où la recherche a été initiée et où elle doit être réalisée, ainsi que des normes et standards internationaux applicables. Les protections garanties par la présente Déclaration aux participants à la recherche ne peuvent être restreintes ou exclues par aucune disposition éthique, légale ou réglementaire, nationale ou internationale.
- 11. La recherche médicale devrait être conçue et menée de manière à éviter ou à réduire les dommages causés à l'environnement, ainsi qu'à encourager la durabilité environnementale.
- 12. La recherche médicale impliquant des participants humains doit être conduite uniquement par des personnes ayant acquis une éducation, une formation et des qualifications appropriées en éthique et en science. Cette recherche nécessite la supervision d'un médecin ou d'un autre chercheur compétent et dûment qualifié. L'intégrité scientifique est essentielle dans la conduite de la recherche médicale impliquant des participants humains. Les personnes, les équipes et les organisations impliquées ne doivent jamais s'engager dans des méconduites en matière de recherche.
- 13. Les groupes sous-représentés dans la recherche médicale devraient bénéficier d'un accès approprié pour participer à la recherche.
- 14. Les médecins qui associent la recherche médicale à des soins médicaux devraient impliquer leurs patients dans une recherche uniquement dans la mesure où elle se justifie par sa valeur potentielle en matière de prévention, de diagnostic ou de traitement et si les médecins ont de bonnes raisons de penser que la participation à la recherche ne portera pas atteinte à la santé des participants concernés.
- 15. Une compensation et un traitement adéquats doivent être garantis pour les participants qui auraient subi un préjudice en raison de leur participation à une recherche.

#### Risques, inconvénients et bénéfices

16. Dans la pratique médicale et la recherche médicale, la plupart des interventions comportent des risques et des inconvénients.

Une recherche médicale impliquant des participants humains ne peut être conduite que si l'importance de l'objectif surpasse les risques et inconvénients pour les participants impliqués.

Version n°2 du 08.10.2025 CONFIDENTIEL Page **49** sur **54** 





17. Toute recherche médicale impliquant des participants humains doit être précédée d'une évaluation minutieuse des risques et des inconvénients prévisibles pour les personnes et les groupes impliqués dans la recherche par rapport aux bénéfices prévisibles pour eux et pour d'autres personnes ou groupes affectés par la pathologie étudiée.

Toutes les mesures destinées à réduire les risques et les inconvénients doivent être mises en œuvre. Les risques et les inconvénients doivent être constamment surveillés, évalués et documentés par le chercheur.

18. Les médecins et les autres chercheurs ne peuvent s'engager dans des recherches impliquant des participants humains que s'ils sont convaincus que les risques et les inconvénients ont été correctement évalués et que ceux-ci peuvent être gérés de manière satisfaisante.

Lorsque les risques et les inconvénients l'emportent sur les bénéfices potentiels ou lorsqu'il existe des preuves concluantes de résultats définitifs, les médecins et les autres chercheurs doivent déterminer s'il convient de poursuivre, de modifier ou de mettre fin immédiatement à la recherche.

#### Vulnérabilité individuelle, collective et communautaire :

- 19. Certaines personnes, certains groupes et certaines communautés se trouvent dans une situation de plus grande vulnérabilité en tant que participants à la recherche, en raison de facteurs qui peuvent être fixes, ou contextuels et dynamiques, et courent ainsi un plus grand risque d'être abusés ou de subir un préjudice. Lorsque ces personnes, groupes et communautés ont des besoins particuliers en matière de santé, leur exclusion de la recherche médicale peut potentiellement perpétuer ou exacerber leurs disparités. Dès lors, les préjudices liés à leur exclusion doivent être pris en compte et mis en balance par rapport aux préjudices liés à leur inclusion. Afin d'être inclus de manière équitable et responsable dans la recherche, ces personnes, groupes et communautés devraient bénéficier d'un soutien et de protections spécifiques.
- 20. La recherche médicale incluant des personnes, groupes ou communautés en situation de vulnérabilité particulière n'est justifiée que si elle répond à leurs besoins et priorités en matière de santé et si la personne, le groupe ou la communauté est susceptible de bénéficier des connaissances, des pratiques ou des interventions qui en résulteront. Les chercheurs ne devraient inclure les personnes en situation de vulnérabilité particulière que si la recherche ne peut être effectuée avec un groupe ou une communauté moins vulnérable, ou si leur exclusion risque de perpétuer ou d'exacerber leurs disparités.

#### Exigences scientifiques et protocoles de recherche

- 21. La recherche médicale impliquant des participants humains doit être conçue et conduite de manière rigoureuse et scientifiquement fondée, afin de produire des connaissances fiables, valides et pertinentes, et d'éviter le gaspillage de la recherche. La recherche doit être conforme aux principes scientifiques généralement acceptés, se baser sur une connaissance approfondie de la littérature scientifique, sur d'autres sources pertinentes d'informations et sur des expériences appropriées en laboratoire et, le cas échéant, sur les animaux. Le bien-être des animaux utilisés dans le cadre de la recherche doit être respecté.
- 22. La conception et la conduite de toute recherche médicale impliquant des participants humains doivent être clairement décrites et justifiées dans un protocole de recherche.

Le protocole devrait contenir une déclaration sur les enjeux éthiques en question et indiquer comment les principes de la présente Déclaration ont été pris en considération. Le protocole devrait inclure des informations sur les objectifs, les méthodes, les bénéfices attendus et les risques et les inconvénients éventuels, les qualifications du chercheur, les sources de financement, les conflits d'intérêts éventuels, les dispositions visant à protéger la vie privée et la confidentialité, les mesures d'incitation pour les participants, les dispositions

Version n°2 du 08.10.2025 CONFIDENTIEL Page **50** sur **54** 





relatives au traitement et/ou à l'indemnisation des participants qui subissent un préjudice en raison de leur participation, et tout autre aspect pertinent de la recherche.

Dans les essais cliniques, le protocole doit aussi décrire toutes les dispositions pour accéder à l'intervention testée après l'essai.

#### Comités d'éthique de la recherche

23. Le protocole doit être soumis pour examen, commentaires, recommandations et approbation au comité d'éthique de la recherche concerné avant le début de la recherche. Ce comité doit fonctionner de manière transparente, et doit disposer de l'indépendance et de l'autorité nécessaires pour résister à toute influence indue de la part du chercheur, du promoteur ou d'autres personnes. Le comité doit disposer de ressources suffisantes pour remplir ses fonctions, et ses membres et son personnel doivent collectivement disposer d'une éducation, d'une formation, de qualifications et d'une diversité adéquates pour évaluer efficacement chaque type de recherche qu'il examine.

Le comité doit avoir une connaissance suffisante des circonstances et du contexte locaux, et comporter au moins un membre du grand public. Il doit prendre en considération les normes et standards éthiques, légaux et réglementaires du ou des pays dans lesquels la recherche doit être menée, ainsi que les normes et standards internationaux applicables, lesquels ne peuvent toutefois restreindre ni exclure aucune des protections garanties aux participants à la recherche par la présente Déclaration.

Lorsqu'une recherche collaborative est menée à l'échelle internationale, le protocole de recherche doit être approuvé par les comités d'éthique de la recherche dans le pays du promoteur et dans les pays hôtes.

Le comité doit avoir le droit de surveiller, de recommander des modifications, de retirer son approbation et de suspendre la recherche en cours. Le chercheur doit fournir des informations au comité et/ou à l'entité compétente en matière de surveillance des données et de sécurité lorsqu'une surveillance est requise, et en particulier en cas d'événement indésirable grave. Aucun amendement ne peut être apporté au protocole sans l'examen et l'approbation du comité. Une fois la recherche terminée, les chercheurs doivent soumettre un rapport final au comité contenant un résumé des résultats et des conclusions.

#### Vie privée et confidentialité

24. Toutes les précautions doivent être prises pour protéger la vie privée des participants à la recherche et la confidentialité de leurs informations personnelles.

#### Consentement libre et éclairé

- 25. Le consentement libre et éclairé est une composante essentielle du respect de l'autonomie individuelle. La participation à la recherche médicale de personnes capables de donner leur consentement éclairé doit être volontaire. Bien qu'il puisse être approprié de consulter les membres de leur famille ou des représentants de leur communauté, les personnes capables de donner leur consentement éclairé ne peuvent être incluses dans une recherche que si elles y consentent librement.
- 26. Dans la recherche médicale impliquant des participants humains capables de donner leur consentement éclairé, chaque participant potentiel doit être informé de manière adéquate et dans un langage courant des objectifs, des méthodes, des bénéfices attendus, des risques et des inconvénients éventuels, des qualifications du chercheur, des sources de financement, des conflits d'intérêts éventuels, des dispositions visant à protéger la vie privée et la confidentialité, des mesures d'incitation pour les participants, des dispositions relatives au traitement et/ou à l'indemnisation des participants qui subissent un préjudice en raison de leur participation, et de tout autre aspect pertinent de la recherche.

Le participant potentiel doit être informé de son droit de refuser de participer à la recherche et de retirer son consentement à participer à tout moment sans subir des mesures de rétorsion. Une attention particulière doit être

Version n°2 du 08.10.2025 CONFIDENTIEL Page **51** sur **54** 





accordée aux besoins spécifiques en matière d'information et de communication de chaque participant potentiel, ainsi qu'aux méthodes utilisées pour transmettre les informations.

Après s'être assuré que le participant potentiel a compris les informations, le médecin ou une autre personne qualifiée doit ensuite obtenir son consentement libre et éclairé, formellement documenté sur papier ou par voie électronique. Si le consentement ne peut pas être exprimé sur papier ou par voie électronique, un consentement non écrit doit être formellement attesté et documenté.

Tous les participants à la recherche médicale devraient avoir le choix d'être informés des conclusions générales et des résultats de la recherche.

- 27. Lorsqu'il cherche à obtenir un consentement éclairé pour participer à une recherche, le médecin ou un autre chercheur doit être particulièrement attentif au cas où le participant potentiel est dans une relation de dépendance avec lui ou pourrait donner son consentement sous la contrainte. Dans ce cas, le consentement éclairé doit être sollicité par une personne qualifiée en la matière et complètement indépendante de cette relation.
- 28. Dans la recherche médicale impliquant des participants humains incapables de donner leur consentement libre et éclairé, le médecin ou une autre personne qualifiée doit solliciter le consentement éclairé du représentant légal, en tenant compte des préférences et des valeurs exprimées par le participant potentiel.

Les personnes incapables de donner leur consentement libre et éclairé se trouvent dans une situation de vulnérabilité particulière et ont droit aux garanties correspondantes. En plus de bénéficier des protections prévues pour les personnes particulièrement vulnérables, les personnes incapables de donner leur consentement ne doivent être incluses dans la rechercher que si celle-ci est susceptible de leur apporter un bénéfice personnel ou si elle n'entraîne que des risques et des inconvénients minimes.

- 29. Lorsqu'un participant potentiel à la recherche qui est incapable de donner son consentement libre et éclairé est en mesure de donner son assentiment aux décisions relatives à sa participation à la recherche, le médecin ou une autre personne qualifiée doit obtenir cet assentiment en plus du consentement du représentant légal autorisé, en tenant compte des préférences et des valeurs exprimées par le participant potentiel. Le désaccord du participant potentiel devrait être respecté.
- 30. La recherche impliquant des participants physiquement ou mentalement incapables de donner leur consentement (par exemple, des patients inconscients) ne peut être menée que si l'état physique ou mental qui empêche de donner un consentement éclairé constitue une caractéristique nécessaire du groupe sur lequel porte cette recherche. Dans de telles circonstances, le médecin ou une autre personne qualifiée doit solliciter le consentement éclairé du représentant légal. Si aucun représentant n'est disponible et que la recherche ne peut pas être retardée, celle-ci peut se poursuivre sans consentement éclairé, à condition que le protocole de recherche mentionne les raisons spécifiques d'impliquer des participants dont l'état les rend incapables de donner leur consentement éclairé et que la recherche ait été approuvée par un comité d'éthique de la recherche.

Le consentement libre et éclairé à participer à la recherche doit être obtenu dès que possible auprès d'un représentant légal ou du participant, si celui-ci recouvre la capacité de donner son consentement.

- 31. Le médecin ou un autre chercheur doit informer pleinement les participants potentiels des aspects de leurs soins qui sont liés à la recherche. Le refus d'un patient de participer à la recherche ou sa décision de se retirer de la recherche ne doit jamais affecter négativement la relation patient/médecin ou la qualité des soins.
- 32. Les médecins ou d'autres personnes qualifiées doivent obtenir le consentement libre et éclairé des participants à la recherche pour le recueil, le traitement, la conservation et l'utilisation secondaire prévisible de matériel biologique et de données identifiables ou ré-identifiables. Toute collecte et conservation de données ou

Version n°2 du 08.10.2025 CONFIDENTIEL Page **52** sur **54** 





de matériel biologique provenant de participants à la recherche pour des utilisations multiples et indéfinies doivent être conformes aux exigences énoncées dans la Déclaration de Taipei de l'AMM, y compris les droits des personnes et les principes de gouvernance. Un comité d'éthique de la recherche doit approuver la création et surveiller l'utilisation continue de ces bases de données et biobanques.

Lorsqu'il est impossible ou irréalisable d'obtenir le consentement, la recherche secondaire sur les données ou le matériel biologique conservés ne peut être effectuée qu'après examen et approbation d'un comité d'éthique de la recherche.

#### <u>Utilisation de placebo</u>

- 33. Les bénéfices, les risques, les inconvénients, ainsi que l'efficacité d'une nouvelle intervention doivent être comparés à ceux de la ou des meilleures interventions éprouvées, sauf dans les circonstances suivantes :
  - S'il n'existe pas d'intervention éprouvées, l'utilisation d'un placebo ou l'absence d'intervention est acceptable ;
  - Si, pour des raisons méthodologiques convaincantes et scientifiquement valables, la réalisation d'une intervention autre que la ou les meilleures éprouvées, l'utilisation d'un placebo ou l'absence d'intervention est nécessaire pour déterminer l'efficacité ou la sécurité d'une intervention, et si les participants qui bénéficient d'une intervention autre que la ou les meilleures éprouvées, d'un placebo ou ne bénéficient d'aucune intervention ne sont pas exposés à des risques supplémentaires de préjudices graves ou irréversibles du fait qu'ils n'ont pas bénéficié de la meilleure intervention éprouvée.

Le plus grand soin doit être apporté afin d'éviter tout abus de cette option.

#### Accès à l'intervention testée après un essai clinique

34. Avant un essai clinique, les promoteurs et les chercheurs doivent prendre des dispositions afin que les participants qui ont encore besoin d'une intervention jugée bénéfique et raisonnablement sûre dans le cadre de l'essai puissent continuer à en bénéficier et que celle-ci soit prise en charge par eux-mêmes, par les systèmes de soins ou par les pouvoirs publics. Les exceptions à cette exigence doivent être approuvées par un comité d'éthique de la recherche. Des informations spécifiques concernant l'accès à l'intervention testée après l'essai clinique doivent être communiquées aux participants dans le cadre du consentement éclairé.

#### Enregistrement des recherches, publication et diffusion des résultats

- 35. Toute recherche médicale impliquant des participants humains doit être enregistrée dans une base de données accessible au public avant le recrutement du premier participant.
- 36. Les chercheurs, auteurs, promoteurs, rédacteurs et éditeurs ont tous des obligations éthiques concernant la publication et la diffusion des résultats de la recherche. Les chercheurs ont le devoir de mettre à la disposition du public les résultats de leurs recherches impliquant des participants humains et ont la responsabilité de fournir leurs rapports de manière rapide, exhaustive et précise. Toutes les parties devraient se conformer aux directives acceptées en matière d'éthique pour la rédaction de rapports. Les résultats aussi bien négatifs et non concluants que positifs doivent être publiés ou rendus publics par un autre moyen. La publication doit mentionner les sources de financement, les affiliations institutionnelles et les conflits d'intérêts. Les rapports de recherche non conformes aux principes de la présente Déclaration ne devraient pas être acceptés pour publication.

### Interventions non éprouvées dans la pratique clinique

37. Lorsqu'une intervention non éprouvée est réalisée pour tenter de rétablir la santé ou de soulager la souffrance d'un patient parce que les options approuvées sont inadéquates ou inefficaces et qu'il n'est pas possible pour le patient de participer à un essai clinique, elle doit ensuite faire l'objet d'une recherche visant à

Version n°2 du 08.10.2025 CONFIDENTIEL Page **53** sur **54** 





évaluer sa sécurité et son efficacité. Les médecins qui participent à de telles interventions doivent demander au préalable l'avis d'experts, évaluer les risques, les inconvénients et les bénéfices possibles, et obtenir le consentement éclairé du patient. Ils doivent également enregistrer et partager les données de manière adéquate et éviter de compromettre les essais cliniques. Ces interventions ne doivent jamais être réalisées pour contourner les protections des participants à la recherche énoncées dans la présente Déclaration.

Version n°2 du 08.10.2025 CONFIDENTIEL Page **54** sur **54**